### **Table of Contents**

| Table of Contents | 3 |
|------------------------------------------------------|----|
| List of Abbreviations and Definitions of Terms | 4 |
| 1. INTRODUCTION | 5 |
| 2. STUDY OBJECTIVES | 5 |
| 3. STUDY DESIGN | 5 |
| 4. HARDWARE AND SOFTWARE | 7 |
| 5. STATISTICAL DATA REVIEW | 8 |
| 6. DATABASE CLOSURE | 8 |
| 7. SAMPLE SIZE DETERMINATION | 8 |
| 8. HANDLING OF MISSING DATA | 8 |
| 9. ANALYSIS POPULATIONS | 8 |
| 10. STATISTICAL EVALUATION | 9 |
| 10.1 Subject Disposition | 9 |
| 10.2 Demographic and Other Covariates | 9 |
| 10.3 Pharmacokinetics Evaluations | 9 |
| 10.4 Safety Evaluations | 11 |
| 11. CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES | 12 |
| 12. HEADINGS | 12 |
| 13. ARCHIVING AND RETENTION OF DOCUMENTS | 13 |
| 15. OUTLINE OF PROPOSED TABLES, FIGURES AND LISTINGS | 14 |



### STATISTICAL ANALYSIS PLAN

A Phase 1, Drug-Drug Interaction Study to Evaluate the Safety, Tolerability, and the Induction potential of TBAJ-876 on CYP3A4 and P-glycoprotein and the Inhibition potential of TBAJ-876 on P-glycoprotein in Healthy Adult Subjects

> Protocol No: TBAJ-876-CL002 TKL Study Number P1980322

> > TKL Research, Inc One Promenade Blvd Fair Lawn, NJ 07410

Jerry Nedelman Senior Director, Pharmacometrics TB Alliance

Michael Tuley, PhD Vice President, Data Sciences and Quality Assurance TKL Research, Inc.

DocuSigned by:

Signer Name: Jerry Nedelman
Signing Reason: I have reviewed the document 22
Signing Time: 12/16/2022 | 8:01:50 AM PST
Signature
DocuSigned by:

Michael Tuley
Signing Reason: I approve this document 2/16/2022
Signing Time: 12/16/2022 | 8:01:37 AM PST
Signing Time: 12/16/2022 | 8:01:37 AM PST
Signing Time: 12/16/2022 | 8:01:37 AM PST
Signing Time: 12/16/2022 | 8:01:37 AM PST
Signing Time: 12/16/2022 | 8:01:37 AM PST
Signing Time: 12/16/2022 | 8:01:37 AM PST

### **Table of Contents**

| 13. | ARCHIVING AND RETENTION OF DOCUMENTS | 12 |
|------|------------------------------------------------|----|
| 12. | HEADINGS | 11 |
| 11. | CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES | 11 |
| | 10.4 Safety Evaluations | 10 |
| | 10.3 Pharmacokinetics Evaluations | 8 |
| | 10.2 Demographic and Other Covariates | 8 |
| | 10.1 Subject Disposition | 8 |
| 10. | STATISTICAL EVALUATION | 8 |
| 9. | ANALYSIS POPULATIONS | 7 |
| 8. | HANDLING OF MISSING DATA | 7 |
| 7. | SAMPLE SIZE DETERMINATION | 7 |
| 6. | DATABASE CLOSURE | 7 |
| 5. | STATISTICAL DATA REVIEW | 7 |
| 4. | HARDWARE AND SOFTWARE | 6 |
| 3. | STUDY DESIGN | 4 |
| 2. | STUDY OBJECTIVES | 4 |
| 1. | INTRODUCTION | 4 |
| List | t of Abbreviations and Definitions of Terms | |
| | ole of Contents | |
| TT - | | _ |

### **List of Abbreviations and Definitions of Terms**

| Abbreviation | Definition |
|--------------|----------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ANOVA | Analysis of variance |
| AUC | Area under the curve |
| CI | Confidence interval |
| CRF | Case Report Form |
| DMP | Data Management Plan |
| ECG | Electrocardiogram |
| ET | Early termination |
| GMR | Ratio of geometric means |
| ODS | Output Delivery System |
| PK | Pharmacokinetics |
| PT | Preferred Term |
| RTF | Rich-Text Format |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TEAE | Treatment-emergent adverse event |

### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the study protocol dated 20 May 2022. This document specifies, in advance of data collection, a comprehensive description of the analysis methods planned to achieve the study objectives specified in the study protocol. Two sequential study phases are planned, with the performance of the second phase conditional on the outcome of the first. The present document will show the planned data presentations, summaries, and analyses for the initial phase of the study. A similar document will be prepared separately in the event that the study enters its second phase.

### 2. STUDY OBJECTIVES

The primary objective of the study is to evaluate the induction potential of TBAJ-876 on CYP3A4 and P-glycoprotein and the inhibition potential of TBAJ-876 on P-glycoprotein in healthy adult subjects.

The secondary objective of the study is to evaluate the effects of multiple-dose administrations of TBAJ-876 on the safety and tolerability of midazolam and digoxin. An extension of the study is planned conditionally on the outcomes of the initial phase, the objective of which will be to evaluate the effects of multiple-dose administration of TBAJ-876 on the safety and tolerability of an antiretroviral regimen.

### 3. STUDY DESIGN

This is a phase 1, open-label, single-center, drug-drug interaction study. Two sequential study phases are planned. The performance of the second phase is conditional on the outcome of the first. The planned enrollment to the first phase of the study is 28 healthy males and females between 18 and 55 years of age. This phase of the study will last 34 days for each subject, from Check-in on Day –1 through completion of the clinical procedures on Day 25 and a follow-up phone call on Day 32.

Subjects will be screened for eligibility to participate in the study up to 21 days prior to admission to the study center on Day –1. Eligible subjects will be admitted to the study center on Day –1 and will be confined there under observation until they are discharged on Day 25. Following discharge, subjects will receive a follow-up phone call on Day 32.

All subjects will receive treatment with single daily doses according to the following schedule:

| Day 1 | Midazolam oral syrup, 2 mg | Fasted |
|---|---|---|
| Day 2 | Digoxin tablet, 0.25 mg | Fasted |
| Day 6 – 13 | TBAJ-876 oral suspension, 200 mg | Fed |
| Day 14 – 19 | TBAJ-876 oral suspension, 165 mg | Fed |
| Day 20 | Midazolam oral syrup, 2 mg; TBAJ-876 oral suspension, 200 mg | Fasted |
| Day 21 | Digoxin tablet, 0.25 mg; TBAJ-876 oral suspension, 200 mg | Fasted |
| Day 22 – 24 | TBAJ-876 oral suspension, 150 mg | Fed |

The following safety assessments will be performed at scheduled time points throughout the study:

| Physical examinations | Screening and Days –1, 2, 3, 4, 5, and 25, or early withdrawal. |
|---|---|
| Vital signs (blood pressure, heart rate [pulse], temperature, and respiration rate, pulse oximetry) | Screening and Days -1 Pre-dose and 0.5, 1, 2, 6, and 12 hours post-dose on Days 1, 2, 6, 20, and 21 6 hours post-dose on Days 7 through 19 Days 24 and 25, or early withdrawal. |
| Electrocardiogram (ECG) | Once at Screening and Days –1, 3, 7, 20, 22, and 25, or upon early withdrawal; also on Days 2 and 21, predose and 0.5, 1, 2, 6, and 12 hours post-dose. |
| Adverse events (AEs) | Ongoing collection throughout the study period. |
| Clinical laboratory tests<br>(hematology, serum chemistry,<br>coagulation, and urinalysis) | Screening and Days –1, 2, 3, 7, 20, 21, 22, and 25, or upon early withdrawal. |

Blood samples will be taken according to the following schedule for determination of plasma concentrations of the corresponding analytes:

| Day 1 | Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours | Midazolam and its metabolite 1-hydroxymidazolam |
|---|---|---|
| Day 2 | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours | Digoxin |
| Day 17 | Pre-dose, 0.5, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24 hours | TBAJ-876 and its metabolites M2 and M3 |
| Day 20 | Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours | Midazolam and its metabolite 1-hydroxymidazolam |
| Day 21 | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours | Digoxin |

### 4. HARDWARE AND SOFTWARE

Statistical analysis will be performed following TKL standard operating procedures (SOPs) and on the TKL computer network. All statistical analyses will be performed using SAS Version 9.4 or higher with program code prepared specifically for the project by qualified TKL statisticians and SAS programmers.

The SAS programs will generate rich-text-formatted (RTF) output with the "RTF" extension using the SAS Output Delivery System (ODS). The summary tables and listings will be formatted using the Times New Roman font. The RTF output is included in report documents prepared with Microsoft Word and converted to PDF format without typographical change.

Study data tabulation model (SDTM) data sets and required analysis data model (ADaM) data sets will be created and taken as input to validated SAS programs to generate the report-ready tables, listings, and figures. Each output display will show the names of the data sets and SAS program used to produce it. Upon completion of the study report, the data sets will be provided to the sponsor as SAS XPT transport files with define.xml files including details of all derivations and imputations used.

### 5. STATISTICAL DATA REVIEW

Data verification activities to be performed prior to delivery of the SAS data sets to the project statistician are described in the approved Data Management Plan (DMP). After completion of the data verification activities, the SAS data sets will be reviewed by the project statistician along with documentation of any unresolved queries and data conventions applied that are not fully explained in the data or in the DMP. The project statistician will perform completeness and self-consistency checks of the study data. These checks will be selected to ensure the self-consistency of dates and events in the subject record, the consistency of all reported data values with expected ranges, and, if not within range, the presence in the subject record of explanatory comments or other corroborative data. Overall, each subject's record in the study database must convey a full but concise description of the subject's experience with respect to protocol-specific events. Questions will be issued to the Data Manager and resolved before closure of the database.

### 6. DATABASE CLOSURE

After completion of all data review procedures, validation of the project database (ie, all those activities and operations designed and performed to ensure that the database is a complete and accurate representation of protocol-specific events), and approval of the data review document by the study sponsor, the clinical database will be closed (ie, "locked"). Any change to the clinical database after this time will require written authorization, with explanation, by the Sponsor and the Biostatistician, in conformance with TKL SOPs.

### 7. SAMPLE SIZE DETERMINATION

The study sample size for this Phase 1 study is based on statistical power calculations as detailed in the study protocol, section 10.2.

### 8. HANDLING OF MISSING DATA

In this study, there will be no imputations of missing data points. All data will be reported and analyzed as observed values only.

### 9. ANALYSIS POPULATIONS

The analysis populations will be determined according to available data. Relevant data for all subjects enrolled to the study will be reported. The Safety population for analysis of adverse events, clinical laboratory test results, and other safety-related variables will include all

subjects who received treatment with any one of the study drugs. The Pharmacokinetics (PK) population for analysis of plasma concentration data and pharmacokinetic parameters will include all subjects presenting data sufficient to calculate the analysis parameter. In case a subject cannot be included in a particular analysis, the rationale for the omission of that subject will be fully explained in the study report.

### 10. STATISTICAL EVALUATION

### 10.1 Subject Disposition

Subject disposition will be summarized by showing the number of subjects screened, and the number and percent of screen failures and enrolled subjects; the number and percent of subjects completed and discontinued, along with the primary reason for discontinuation. By-subject listings will include date of informed consent, date of screening, date-time of enrollment, date of last visit, date of last contact, and reason for discontinuation. Individual subject data for any protocol deviations will also be presented in a by-subject listing.

### 10.2 Demographic and Other Covariates

Subject age, height, weight, and BMI will be summarized for the Safety population as mean, standard deviation, median, minimum, and maximum. Sex, race, and ethnicity will be summarized as number and percent of subjects in each category. Subject listings will include age, sex, race, ethnicity, weight, height, and body mass index.

Prior (prior to the start of treatment) medication use and concomitant (after the start of treatment) medication use will be summarized separately. If the end date of a prior medication occurs after treatment starts, then the medication will be reported in both the prior and concomitant tables and listings. These tables will present the number and percentage of subjects for each medication. Medication terms will be coded and classified according to the WHO Drug Dictionary, Version B3 (March 2022).

Data listings will also be provided to show medical history, childbearing potential and pregnancy test results, and general investigator comments.

### **10.3** Pharmacokinetics Evaluations

Plasma concentrations will be summarized at each time point for each measured analyte as mean, standard deviation, median, coefficient of variation, standard error of the mean, minimum and maximum. Individual subject data will be plotted against time post-dose on linear and log-linear axes. Day 1 and Day 20 midazolam concentrations, and Day 2 and

Day 21 digoxin concentrations, will be overlayed on a single set of axes to permit visual comparison. Similar displays will be constructed for the mean concentrations of each analyte over time post-dose.

The following pharmacokinetics parameters will be determined for each subject and study day for midazolam, 1-hydroxymidazolam, and digoxin:

- AUC<sub>0-last</sub>, the area under the curve of plasma concentration vs time post-dose, approximated trapezoidally, from 0 to the time of last measurable concentration;
- C<sub>max</sub>, the maximum observed concentration;
- $t_{max}$ , the time post-dose of the maximum observed concentration.

The individual subject plots of each analyte concentration vs time will be inspected visually to identify log-linear terminal segments corresponding to an exponential elimination phase. If at least 3 observations are presented along what appears to be a terminal elimination phase, then the elimination rate constant will be estimated using a linear regression fit to the plot of log concentration vs time during this phase. The value of the elimination rate constant, kel, is the absolute magnitude of the estimated slope.

Using the following SAS code,

the value of  $k_{el}$  is computed as ABS(TIME) in the dataset KOUT, and the value of the elimination half-life,  $t_{1/2}$ , is LOG(2)/KEL.

When  $k_{el}$  and  $t_{1/2}$  are estimated, the following additional parameters will be computed:

- AUC<sub>0-inf</sub>, the area under the curve of plasma concentration vs time post-dose, extrapolated to infinite time, calculated as  $AUC_{0-last} + C_{last}/k_{el}$ ;
- CL/F, total apparent drug clearance rate, defined as oral dose / AUC<sub>0-inf</sub>; (Note that when oral dose is provided in units of mg, the AUC must be converted to units of mg.hr/L.)
- V<sub>Z</sub>/F, apparent volume of distribution, defined as CL/F divided by k<sub>el</sub>.

In addition to mean, standard deviation, median, minimum, and maximum, the AUC parameters and Cmax will be summarized by treatment group as geometric mean and coefficient of variation (ie, 100\*SQRT(EXP(VAR) - 1) with VAR= the variance of the log-

transformed values). Elimination rate constant, half-life, and t<sub>max</sub> will be summarized as median, minimum, and maximum. Drug clearance and volume of distribution will be summarized as mean, standard deviation, minimum, and maximum.

To compare pharmacokinetic parameters of the interaction products with TBAJ-876 versus alone, analyses of variance (ANOVA) will be performed using SAS PROC MIXED. The model will include subject as a random effect and treatment (with TBAJ-876 versus alone) as a fixed effect. Geometric least-squares mean values and 95% confidence intervals (CIs) will be tabulated for AUC<sub>0-inf</sub> and C<sub>max</sub>. The ratio of geometric means (GMR) will be computed comparing co-administration with TBAJ-876 versus alone, along with the 90% 2-sided CI. The test drug TBAJ-876 will be considered a moderate inducer of CYP3A4 if the estimated GMR of midazolam AUC<sub>0-inf</sub> is less than 0.50. It will be considered a moderate inducer of P-glycoprotein if the estimated GMR of digoxin AUC<sub>0-inf</sub> is less than 0.50. If the estimated GMR of digoxin AUC<sub>0-inf</sub> is 2.0 or greater, then TBAJ-876 will be considered a moderate inhibitor of P-glycoprotein. These results will be used to decide whether to conduct the second phase of the study.

The following pharmacokinetics parameters will be determined for each subject for TBAJ-876 and its metabolites M2 and M3 on Day 17:

- AUC<sub>0-24</sub>, the area under the curve of plasma concentration vs time post-dose, approximated trapezoidally, from 0 to 24 hours post-dose;
- C<sub>max</sub>, the maximum observed concentration;
- $t_{max}$ , the time post-dose of the maximum observed concentration.
- C<sub>trough</sub>, the observed pre-dose concentration.

The sum of AUC<sub>0-24</sub> for TBAJ-876 and its M3 metabolite will also be summarized. In addition to mean, standard deviation, median, minimum, and maximum, the AUC parameters and Cmax will be summarized by treatment group as geometric mean and coefficient of variation (ie, 100\*SQRT( EXP(VAR) - 1 ) with VAR= the variance of the log-transformed values). The summary of t<sub>max</sub> will be as median, minimum, and maximum. Trough concentration will be summarized as mean, standard deviation, minimum, and maximum.

### **10.4** Safety Evaluations

All safety analysis will be performed using the Safety analysis population and will be presented by group Adverse event terms will be coded using the MedDRA version 25 (2022) dictionary. All AEs will be presented in a by-subject listing, detailing the verbatim term given by the investigator, the preferred term (PT), system organ class (SOC), onset date and time, end date

and time, severity, outcome, relationship to study drug, action taken with study drug, other action taken, seriousness and criteria for seriousness.

All safety and tolerability data collected in the study will be listed by participant. The continuous variables will be summarized using number of eligible subjects (N), mean, standard deviation, median, minimum, and maximum. Frequency counts and percentages will be reported for categorical data.

A treatment emergent adverse event is defined as an AE beginning on or after Day 1 of the study. The number of events and the number and percent of subjects experiencing adverse events will be presented for all treatment-emergent adverse events (TEAE), all treatment-related TEAEs, all severe TEAEs (Grades 3 and 4), and all TEAEs leading to study discontinuation. Number and percent of subjects with TEAEs will also be shown by SOC and PT.

Vital signs, ECG measurements, and clinical laboratory test results (including hematology, serum chemistry, coagulation, and urinalysis) will be summarized at each time point as mean, standard deviation, median, minimum, and maximum. The investigator's assessments of ECG as normal or abnormal will be summarized as number and percentage of subjects. Also, the presence of heart murmur at each time point will be summarized as number and percentage of subjects. Every cardiovascular safety incident will be listed by timepoint with accompanying symptoms and with BP and HR measurements.

The results of all safety-related data, including physical examinations findings, vital signs, ECG assessments, and clinical laboratory test results, will be presented in by-subject listings.

### 11. CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES

All exceptions to the planned analyses as described herein will be clearly indicated and explained in the study report.

### 12. HEADINGS

Each page of the analysis will show the sponsor's name, the investigational product, and the protocol number. Report tables will be embedded in the MS Word report document from SAS program output without change. The footer of each table will show the name of the SAS program module which generated it, the names of all data sets providing input data in the program and the date and time the table was generated.

### 13. ARCHIVING AND RETENTION OF DOCUMENTS

After finalization of the analysis, the following will be archived at TKL Research, Inc. and/or with the study sponsor:

- SAP and any amendments
- DMP and Database Specification
- All SAS code used in the project for statistical analysis, report tables generation, and analysis data set creation
- Tables, listings and figures as included in the clinical study report
- SDTM and ADaM datasets
- Relevant correspondence
- Any other pertinent study document (ie, study protocol, investigator's brochure, correspondence, study report, etc.).

# 15. OUTLINE OF PROPOSED TABLES, FIGURES AND LISTINGS

# **Summary Tables**

| 14.1.1 | Summary of Subject Disposition |
|---|---|
| 14.1.2 | Summary of Subject Demographics and Baseline Variables |
| 14.1.3 | Summary of Prior Medications |
| 14.1.4 | Summary of Concomitant Medications |
| 14.2.1.1 | Summary of Plasma Midazolam Concentrations (ng/mL) |
| 14.2.1.2 | Summary of Plasma Digoxin Concentrations (ng/mL) |
| 14.2.1.3 | Summary of Day 17 Plasma TBAJ-876 Concentrations (ng/mL) |
| 14.2.2 | Summary of Drug-Drug Interaction |
| 14.2.3.1 | Summary of Midazolam Pharmacokinetic Parameters |
| 14.2.3.2 | Summary of Digoxin Pharmacokinetic Parameters |
| 14.2.3.3 | Summary of Day 17 TBAJ-876 Pharmacokinetic Parameters |
| 14.3.1 | Summary of Treatment-Emergent Adverse Events |
| 14.3.2 | Summary of Physical Examinations Findings |
| 14.3.3 | Summary of Vital Signs |
| 14.3.4 | Summary of ECG Findings |
| 14.3.5.1 | Summary of Clinical Laboratory Test Results, Hematology and Coagulation |
| 14.3.5.2 | Summary of Clinical Laboratory Test Results, Differential Blood Count |
| 14.3.5.3 | Summary of Clinical Laboratory Test Results, Electrolytes and Renal Function |
| 14.3.5.4 | Summary of Clinical Laboratory Test Results, Liver Function |
| 14.3.5.5 | Summary of Clinical Laboratory Test Results, Other Serum Chemistry |
| 14.3.5.6 | Summary of Clinical Laboratory Test Results, Urinalysis, Part 1 |
| 14.3.5.7 | Summary of Clinical Laboratory Test Results, Urinalysis, Part 2 |

## Figures

| 14.2.1 | Mean Plasma Midazolam Concentration vs Time Post-dose |
|---|---|
| 14.2.2 | Mean Plasma 1-Hydroxymidazolam Concentration vs Time Post-dose |
| 14.2.3 | Mean Plasma Digoxin Concentration vs Time Post-dose |
| 14.2.4 | Mean Day 17 Plasma TBAJ-876 Concentration vs Time Post-dose |
| 14.2.5 | Mean Day 17 Plasma M2 Concentration vs Time Post-dose |
| 14.2.6 | Mean Day 17 Plasma M3 Concentration vs Time Post-dose |
| 14.3.1.1 | Individual Subjects Plasma Midazolam Concentration vs Time Post-dose, Linear Scale |
| 14.3.1.2 | Individual Subjects Plasma Midazolam Concentration vs Time Post-dose, Log-linear Scale |
| 14.3.2.1 | Individual Subjects Plasma 1-Hydroxymidazolam Concentration vs Time Post-dose, Linear Scale |
| 14.3.2.2 | Individual Subjects Plasma 1-Hydroxymidazolam Concentration vs Time Post-dose, Log-linear Scale |
| 14.3.3.1 | Individual Subjects Plasma Digoxin Concentration vs Time Post-dose, Linear Scale |
| 14.3.3.2 | Individual Subjects Plasma Digoxin Concentration vs Time Post-dose, Log-linear Scale |
| 14.3.4 | Individual Subjects Day 17 Plasma TBAJ-876 Concentration vs Time Post-dose |
| 14.3.5 | Individual Subjects Day 17 Plasma M2 Concentration vs Time Post-dose |
| 14.3.6 | Individual Subjects Day 17 Plasma M3 Concentration vs Time Post-dose |

# Listings

| 16.1.7 | Subject Enrollment |
|----------|-------------------------------------------|
| 16.2.1.1 | Screen Failures |
| 16.2.1.2 | Subject Disposition |
| 16.2.2 | Protocol Deviations |
| 16.2.4.1 | Demographics and Baseline Characteristics |
| 16.2.4.2 | Prior and Concomitant Medication |
| 16.2.4.3 | Medical History |

| 16.2.5.1 | Plasma Midazolam Concentrations |
|---|---|
| 16.2.5.2 | Plasma 1-Hydroxymidazolam Concentrations |
| 16.2.5.3 | Plasma Digoxin Concentrations |
| 16.2.5.4 | Plasma TBAJ-876 Concentrations |
| 16.2.5.5 | Plasma M2 Concentrations |
| 16.2.5.6 | Plasma M3 Concentrations |
| 16.2.6.1 | Midazolam Pharmacokinetic Parameters |
| 16.2.6.2 | 1-Hydroxymidazolam Pharmacokinetic Parameters |
| 16.2.6.3 | Digoxin Pharmacokinetic Parameters |
| 16.2.6.4 | TBAJ-876 Dosing |
| 16.2.6.5 | TBAJ-876 Day 17 Pharmacokinetic Parameters |
| 16.2.7.1 | Adverse Events |
| 16.2.7.2 | Serious Adverse Events and Adverse Events Leading to Study Discontinuation |
| 16.2.7.3 | Cardiovascular Adverse Events |
| 16.2.8.1 | Physical Examinations |
| 16.2.8.2 | Vital Signs Measurements |
| 16.2.8.3 | Electrocardiogram (ECG) Results |
| 16.2.8.4.1 | Clinical Laboratory Test Results, Hematology and Coagulation |
| 16.2.8.4.2 | Clinical Laboratory Test Results, Differential Blood Count |
| 16.2.8.4.3 | Clinical Laboratory Test Results, Electrolytes and Renal Function |
| 16.2.8.4.4 | Clinical Laboratory Test Results, Liver Function |
| 16.2.8.4.5 | Clinical Laboratory Test Results, Other Serum Chemistry |
| 16.2.8.4.6 | Clinical Laboratory Test Results, Urinalysis, Part 1 |
| 16.2.8.4.7 | Clinical Laboratory Test Results, Urinalysis, Part 2 |
| 16.2.8.4.8 | Laboratory Values Outside of Normal Range |
| 16.2.8.5 | Childbearing Potential and Serum Pregnancy Test Results |
| 16.2.9 | General Comments |

| Number of Subjects Screened | XX |
|---------------------------------------------------------|-----------|
| n (%) Enrolled | XX (XX.X) |
| n (%) Screen Failure | xx (xx.x) |
| Number Enrolled | XX |
| n (%) Completed Study | xx (xx.x) |
| n (%) Discontinued Study | XX (XX.X) |
| n (%) Adverse Event/Serious Adverse Event | XX (XX.X) |
| n (%) Important Protocol Deviation (eg, non-compliance) | XX (XX.X) |
| n (%) Investigator Judgment | XX (XX.X) |
| n (%) Lost to Follow-up | XX (XX.X) |
| n (%) n xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) |

[Programming Note: List reasons for discontinuation in descending order of frequency. Omit rows with zero counts.]

TB Alliance Protocol No. TBAJ-876-CL002 TKL No. P1980322

| TB Alliance Protocol Number: TBAJ-876-CL002 | 02 | | |
|---|---|---|---|
| | | Table 14.1.2: Summary of Subject Demographics and Baseline Variables Safety population (N=xx) | ariables |
| Par | Parameter | Statistic | |
| Age | v | Mean (SD) | XXX (XX.X) |
| | | Median | XXX |
| | | Minimum, maximum | XXX, XXX |
| Sex | ¥ | n (%) Male | x (xx.x) |
| | | n (%) Female | x (xx.x) |
| Race | es<br>es | n (%) White | x (xx.x) |
| | | n (%) Black or African American | x (xx.x) |
| | | n (%) Asian | x (xx.x) |
| | | n (%) American Indian or Alaska Native | x (xx.x) |
| | | n (%) Native Hawaiian or Other Pacific Islander | x (xx.x) |
| Eth | Ethnicity | n (%) Hispanic or Latino | x (xx.x) |
| | | n (%) Not Hispanic or Latino | x (xx.x) |
| Note: Subjects could select more th | han one race and | Note: Subjects could select more than one race and are counted in each race selected. SD=Standard deviation. | |
| Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX | by XXXXX / U | ses: XX | |

[Programming Note: Omit rows with zero counts.]


| TB Alliance Protocol Number: TBAJ-876-CL002 | | |
|---|---|---|
| | Table 14.1.2: Summary of Subject Demographics and Baseline Variables Safety population (N=xx) | seline Variables |
| Parameter | Statistic | |
| Height (cm) | Mean (SD)<br>Median | XXX (XX.X) |
| | Minimum, maximum | XXX, XXX |
| Weight (kg) | Mean (SD)<br>Median<br>Minimum, maximum | XX.X (XX.X) XX.X XX.X, XX.X |
| BMI (kg/m^2) | Mean (SD)<br>Median<br>Minimum, maximum | XX.X (XX.X) XX.X XX.X, XX.X |
| SD=Standard deviation. | | |
| Generated on XX/XX/XX:XXXX by XXXXXX / Uses: XX | / Uses: XX | |

| TB Alliance Protocol Number: TBAJ-876-CL002 | Page X of Y |
|---|---|
| Table 14.1.3: Summary of Prior Medications Safety population (N=xx) | lications |
| Number (%) of Subjects with Any Prior Medication | xx (xx.x) |
| [ATC2] | xx (xx.x) |
| [WHO Preferred Name 1] | XX (XX.X) |
| [WHO Preferred Name 2] | xx (xx.x) |
| [ATC2] | xx (xx.x) |
| [WHO Preferred Name 1] | XX (XX.X) |
| [WHO Preferred Name 2] | xx (xx.x) |
| [ATC2] | xx (xx.x) |
| [WHO Preferred Name 1] | XX (XX.X) |
| [WHO Preferred Name 2] | xx (xx.x) |
| Note: Medications that were continued into the study period are summarized as both prior and concomitant. | ant. |
| Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX | |

[Programming Note: List ATC2 classes and preferred names in descending order of frequency]


| TB Alliance Protocol Number: TBA1-876-CL002 | Page X of Y |
|---|---|
| Table 14.1.4: Summary of Concomitant Medications Safety population (N=xx) | cations |
| Number (%) of Subjects with Any Concomitant Medication | XX (XX.X) |
| [ATC2] | XX (XX.X) |
| [WHO Preferred Name 1] | xx (xx.x) |
| [WHO Preferred Name 2] | XX (XX.X) |
| [ATC2] | XX (XX.X) |
| [WHO Preferred Name 1] | XX (XX.X) |
| [WHO Preferred Name 2] | XX (XX.X) |
| [ATC2] | XX (XX.X) |
| [WHO Preferred Name 1] | XX (XX.X) |
| [WHO Preferred Name 2] | xx (xx.x) |
| Note: Medications that were continued into the study period are summarized as both prior and concomitant. | |
| Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX | |

[Programming Note: List ATC2 classes and preferred names in descending order of frequency]

Page X of Y

TB Alliance
Protocol Number: TBAJ-876-CL002

Table 14.2.1.1: Summary of Plasma Midazolam Concentrations (ng/mL) PK Population

| | | Mid | Midazolam | 1-Hydrox | 1-Hydroxymidazolam |
|---|---|---|---|---|---|
| Time Point | Statistic | Alone | With TBAJ-876 | Alone | With TBAJ-876 |
| [Pre-dose 15 mins 30 mins 1 hr 2 hrs | | | | | |
| 3 hrs, 4 hrs, 6 hrs, 8 hrs, 12 hrs, 24 hrs] | n | XX | XX | XX | × |
| | Mean (SD) | (X.XX) XXX | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| | Median | XXX | XXX | XXX | XXX |
| | Geometric mean | XXX | XXX | XXX | XXX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |

SD=Standard deviation, CV=Coefficient of variation.


| | ıble 14.2.1.2: Summary of Pl<br>PK | Table 14.2.1.2: Summary of Plasma Digoxin Concentrations (ng/mL) PK Population | (ng/mL) |
|---|---|---|---|
| | | Di | Digoxin |
| Time Point Statistic | stic | Alone | With TBAJ-876 |
| [Pre-dose, 30 mins, 1 hr, 2 hrs, 3 hrs, 4 hrs, 6 hrs, 8 hrs, 12 hrs, 24 hrs, 48 hrs, n 72 hrs, 96 hrs] | | XX | XX |
| | Mean (SD) | XXX (XX.X) | xxx (xx.x) |
| Median | ian | XXX | XXX |
| Geon | Geometric mean | XXX | XXX |
| CV (%) | (%) | XX.X | XX.X |
| Mini | Minimum, maximum | XXX, XXX | XXX, XXX |


| TB Alliance Protocol Number: TBAJ-876-CL002 | | | | Page X of Y |
|---|---|---|---|---|
| | 1 able 14.2.1.3: Summary of Day 17 Plasma 1 BAJ-870 Concentrations (ng/ml.) PK Population | 7 17 Plasma 1 BAJ-870 Concent<br>PK Population | anons (ng/mL) | |
| Time Point | Statistic | TBAJ-876 | M2 | M3 |
| [Pre-dose, 30 mins, 3 hrs, 4 hrs, 5 hrs, 6 hrs, 7 hrs, 8 hrs, 12 hrs, 16 hrs, 20 hrs, 24 hrs] | п | ×× | ×× | xx |
| | Mean (SD) | XXX (XX.X) | XXX(XX.X) | XXX (XX.X) |
| | Median | XXX | XXX | XXX |
| | Geometric mean | XXX | XXX | XXX |
| | CV (%) | XX.X | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX | xxx, xxx |


| TB Alliance Protocol Number: TBAJ-876-CL002 | | Page 1 of 1 |
|---|---|---|
| Table 14.2.2: Summary of Drug-Drug Interaction PK Population | rug-Drug Interaction<br>tion | |
| | Midazolam | Digoxin |
| $\mathrm{AUC}_{O	ext{-}\mathrm{inf}}(\mathrm{ng.hr/mL})$ | N=xx | N=xx |
| Least-squares geometric mean (with TBAJ-876 [T]) | XXX | XXX |
| Least-squares geometric mean (alone [R]) | XXX | XXX |
| Ratio of geometric means (T/R) | X.XXX | X.XXX |
| 90% 2-sided confidence interval | [x.xxx, x.xxx] | [x.xxx, x.xxx] |
| $C_{\max}(ng/mL)$ | N=xx | N=xx<br>N |
| Least-squares geometric mean (with TBAJ-876 [T]) | XXX | XXX |
| Least-squares geometric mean (alone [R]) | XXX | XXX |
| Ratio of geometric means (T/R) | X.XXX | X.XXX |
| 90% 2-sided confidence interval | [x.xxx, x.xxx] | [x.xxx, x.xxx] |

Note: All estimates are of least squares means using the mixed linear model analysis of variance with random effects of subject and fixed effects of treatment.


| TB Alliance Protocol Number: TBAJ-876-CL002 | | | | | ď |
|---|---|---|---|---|---|
| | Table 14.2.3.1: Summary of Midazolam Pharmacokinetic Parameters<br>PK Population | ry of Midazolam Phar<br>PK Population | macokinetic Parameters | | |
| | | Mid | Midazolam | 1-Hydrox | 1-Hydroxymidazolam |
| Parameter | Statistic | Alone | With TBAJ-876 | Alone | With TBAJ-876 |
| AUC <sub>0-last</sub> (ng.hr/mL) | u | XX | XX | XX | × |
| | Mean (SD) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| | Median | XXX | XXX | XXX | XXX |
| | Geometric mean | XXX | XXX | XXX | XXX |
| | CV (%) | XXX.X | XX.X | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| AUC <sub>0-inf</sub> (ng.hr/mL) | и | × | XX | XX | × |
| | Mean (SD) | (X.XX) XXX | XXX(XX.X) | xxx (xx.x) | XXX (XX.X) |
| | Median | XXX | XXX | XXX | XXX |
| | Geometric mean | XXX | XXX | XXX | XXX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| C <sub>max</sub> (ng/mL) | и | XX | ×× | XX | × |
| | Mean (SD) | (x.xx) | (xxx) (xxx) | xxx (xx.x) | XXX (XX.X) |

XX.X XXX, XXX

XX.X XXX, XXX

XX.X XXX, XXX

XX.X XXX, XXX

Median Geometric mean CV (%) Minimum, maximum

XXX XXX

XXX

XXX XXX

XXX XXX


| | | PK Population | PK Population | | |
|---|---|---|---|---|---|
| | | Mid | Midazolam | 1-Hydrox | 1-Hydroxymidazolam |
| Parameter | Statistic | Alone | With TBAJ-876 | Alone | With TBAJ-876 |
| $T_{max}$ (hr) | u | XX | XX | XX | × |
| | Median | XXX | XXX | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| kel (/hr) | и | XX | X | XX | × |
| | Median | XXX | XXX | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| t <sub>1/2</sub> (hr) | и | XX | XX | XX | × |
| | Median | XXX | XXX | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| CL/F (L/hr) | и | XX | ×× | XX | × |
| | Mean (SD) | (X.XX) XXX | XXX(XX.X) | xxx (xx.x) | XXX (XX.X) |
| | Median | XXX | XXX | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| $ m V_Z/F\left(L ight)$ | и | XX | XX | XX | × |
| | Mean (SD) | (x.xx) xxx | XXX(XX.X) | xxx (xx.x) | XXX (XX.X) |
| | Median | XXX | XXX | XXX | XXX |


| TB Alliance Protocol Number: TBAJ-876-CL002 | | | |
|---|---|---|---|
| | Table 14.2.3.2: Summary ( | fable 14.2.3.2: Summary of Digoxin Pharmacokinetic Parameters PK Population | meters |
| | | Di | Digoxin |
| Parameter | Statistic | Alone | With TBAJ-876 |
| AUC <sub>0-last</sub> (ng.hr/mL) | и | XX | XX |
| | Mean (SD) | XXX (XX.X) | XXX (XX.X) |
| | Median | XXX | XXX |
| | Geometric mean | XXX | XXX |
| | CV (%) | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX |
| AUCo-inf (ng.hr/mL) | и | XX | XX |
| | Mean (SD) | xxx (xx.x) | XXX (XX.X) |
| | Median | XXX | XXX |
| | Geometric mean | XXX | XXX |
| | CV (%) | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX |
| $C_{max}$ (ng/mL) | и | X | XX |
| | Mean (SD) | XXX (XX.X) | XXX (XX.X) |
| | Median | XXX | XXX |
| | Geometric mean | XXX | XXX |
| | CV (%) | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX |


| | • | radic 14.2.3.2. Summay of Digorm Fnamiaconnicity Faameers<br>PK Population | |
|---|---|---|---|
| | | Q | Digoxin |
| Parameter | Statistic | Alone | With TBAJ-876 |
| $T_{max}$ (hr) | п | XX | XX |
| | Median | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX |
| kel (/hr) | п | XX | XX |
| | Median | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX |
| t <sub>1/2</sub> (hr) | п | XX | XX |
| | Median | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX |
| CL/F (L/hr) | и | XX | XX |
| | Mean (SD) | XXX (XX.X) | XXX (XX.X) |
| | Median | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX |
| Vz/F (L) | п | XX | XX |
| | Mean (SD) | XXX (XX.X) | XXX (XX.X) |
| | Median | XXX | XXX |


| | Table 14.2.3.3 | Table 14.2.3.3: Summary of Day 17 TBAJ-876 Pharmacokinetic Parameters PK Population | 76 Pharmacokinetic Paramet<br>1 | ers | |
|---|---|---|---|---|---|
| Parameter | | TBAJ-876 | M2 | M3 | Sum of TBAJ-876<br>and M3 |
| AUC <sub>0-24</sub> (ng.hr/mL) | n | XX | XX | XX | XX |
| | Mean (SD) | (X.XX) | XXX (XX.X) | XXX (XX.X) | (X.XX) |
| | Median | XXX | XXX | XXX | XXX |
| | Geometric mean | XXX | XXX | XXX | XXX |
| | CV (%) | XX.X | XX.X | XX.X | XXX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| C <sub>max</sub> (ng/mL) | п | XX | × | × | XX |
| | Mean (SD) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | (X.XX) XXX |
| | Median | XXX | XXX | XXX | XXX |
| | Geometric mean | XXX | XXX | XXX | XXX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| $t_{\max}\left(hr\right)$ | п | XX | XX | XX | XX |
| | Median | XXX | XXX | XXX | XXX |
| | Minimum, maximum | XXX, XXX | XXX, XXX | XXX, XXX | XXX, XXX |
| Ctrough (ng/mL) | n | XX | XX | XX | XX |
| | Mean (SD) | XXX | XXX | XXX | XXX |
| | Minimum maximum | XXX XXX | XXX. XXX | XXX XXX | XXX XXX |


| | Table 14.3.1: Summary of Treatment-Emergent Adverse Events Safety Population (N=xx) | Emergent Adverse Events<br>(N=xx) |
|---|---|---|
| All TEAEs | Number of events<br>n (%) of subjects | XX<br>XX (XX.X) |
| Treatment-related TEAEs | Number of events<br>n (%) of subjects | XX<br>XX (XX.X) |
| Severe TEAEs | Number of events<br>n (%) of subjects | XX<br>XX (XX.X) |
| TEAEs leading to study discontinuation | Number of events<br>n (%) of subjects | XX<br>XX (XX.X) |
| [SOCI] [PTI] [PT2] [PT3] | n (%) of subjects | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| [SOC2] [PT1] [PT2] | | XX (XX.X) XX (XX.X) XX (XX.X) |

TEAE=Treatment-emergent adverse event (with onset on or after Day 1).

| TB Alliance Protocol Number: TBAJ-876-CL002 Table 14.3.2: Summary of Physical Examinations Findings Safety Population |
|---|
|---|

| | | | | | u | n(%) Abnormal | lı | | | | Presence of |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Z | HEENT | Neck | Heart | Resp | Abd | MS | Neur | Skin | Other | Heart<br>Murmur |
| Screening | XX | x (xx.x) | 0 | 0 | 0 | 0 | X (XX.X) | 0 | 0 | 0 | 0 |
| Day -1 | XX | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Day 2 | XX | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Day 3 | XX | 0 | x (xx.x) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Day 4 | XX | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | x (xx.x) |
| Day 5 | XX | 0 | 0 | 0 | 0 | 0 | 0 | 0 | x (xx.x) | 0 | 0 |
| Day 25/ET | XX | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

Resp=Respiratory, Abd=Abdomen, MS=Musculoskeletal, Neur=Neurological status.

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

[Note: Show 0 without percentage as shown.]

| TP Alliance | | | | | | | | | Dogs Vof V |
|---|---|---|---|---|---|---|---|---|---|
| Protocol Number: TBAJ-876-CL002 | 20 | | | | | | | | rage Au i |
| | | | Table 14.3.3: Summary of Vital Signs | ımmary of Vi | tal Signs | | | | |
| | | | Safety | Safety Population | | | | | |
| | Supine | | Supine Supine Heart | | | | Supine | Supine | Supine Heart |
| | Systolic BP | Dig | Rate | Temp | Resp Rate | Resp Rate Pulse Systolic BP Diastolic BP Rate | Systolic BP | Diastolic BP | Rate |
| Time Point | (mmHa) | (mmHa) | (hnm) | ( | (hnm) | Oximetry (%) | (mmHa) | (mmHa) | (hnm) |

| Time Point | | Supine<br>Systolic BP<br>(mmHg) | Supine<br>Diastolic BP<br>(mmHg) | Supine Heart<br>Rate<br>(bpm) | Temp<br>(C) | Resp Rate (bpm) | Pulse<br>Oximetry (%) | Supine<br>Systolic BP<br>(mmHg) | Supine<br>Diastolic BP<br>(mmHg) | Supine Heart<br>Rate<br>(bpm) |
|---|---|---|---|---|---|---|---|---|---|---|
| Screening | ٤ | * | * | * | * | × | ** | * | ** | * |
| Scicening | (49) | v · | v. | vv 、 | vv 、 | vv 、 | vv | v 、 | v | vv |
| | Mean (SD) | XXX (XX.X) | (XXX) XXX | XXX (XX.X) | (X.XX) X.XX | XX.X (XX.X) | XX.X (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| | Median | XXX | XXX | XXX | XX.X | XX.X | XXXX | XXX | XXX | XXX |
| | Min, Max | XXX, XXX | XXX, XXX | XXX, XXX | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XXX, XXX | XXX, XXX | XXX, XXX |
| Day -1 | n | XX | XX | XX | xx | xx | xx | XX | xx | XX |
| | Mean (SD) | xxx (xx.x) | (x.xx) xxx | xxx (xx.x) | (x.x.) x.xx | xx.x (xx.x) | (x.xx) x.xx | xxx (xx.x) | (x.xx) xxx | xxx (xx.x) |
| | Median | xxx | xxx | XXX | X.X.X | x.x.x | XXXX | XXX | XXX | XXX |
| | Min, Max | XXX, XXX | XXX, XXX | XXX, XXX | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XXX, XXX | XXX, XXX | XXX, XXX |
| Day 1, Pre-dose | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xxx (xx.x) | (x.xx) xxx | xxx (xx.x) | xx.x (xx.x) | xx.x (xx.x) | (x.xx) x.xx | xxx (xx.x) | (x.xx) xxx | xxx (xx.x) |
| | Median | XXX | XXX | XXX | X.XX | X.X.X | XXX.X | XXX | xxx | xxx |
| | Min, Max | XXX, XXX | XXX, XXX | XXX, XXX | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XXX, XXX | XXX, XXX | XXX, XXX |
| Day 1, 0.5 hrs | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xxx) | xx.x (xx.x) | (x.xx) x.xx | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Median | XXX | XXX | XXX | X.XX | XX.X | XX.X | XXX | XXX | XXX |
| | Min, Max | XXX, XXX | xxx, xxx | xxx, xxx | xx.x, xx.x | XXX, XXX | XX.X, XX.X | xxx, xxx | xxx, xxx | xxx, xxx |
| etc. | | | | | | | | | | |


| | | | | Table 14.3.4.1: \$<br>Saf | Table 14.3.4.1: Summary of ECG Findings<br>Safety Population | G Findings | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | | HR<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF<br>(msec) | Investigator's Assessment | ssessment |
| Screening | п | XX | XX | XX | XX | XX | | |
| | Mean (SD) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xx.x (xx.x) | XX.X (XX.X) | Normal, n(%) | xx (xx.x) |
| | Median | XXX | XXX | XXX | XXX.X | XX.X | Abnormal, n(%) | xx (xx.x) |
| | Min, Max | XXX, XXX | XXX, XXX | XXX, XXX | XX.X, XX.X | XX.X, XX.X | | |
| Day -1 | n | XX | XX | XX | XX | XX | | |
| | Mean (SD) | xxx (xx.x) | (x.xx) xxx | xxx (xx.x) | XX.X (XX.X) | XX.X (XX.X) | Normal, n(%) | XX (XX.X) |
| | Median | XXX | XXX | XXX | XX.X | XX.X | Abnormal, n(%) | XX (XX.X) |
| | Min, Max | XXX, XXX | XXX, XXX | XXX, XXX | XX.X, XX.X | XX.X, XX.X | | |
| Day 2, Pre-dose | u | X | XX | XX | XX | XX | | |
| | Mean (SD) | XXX (XX.X) | (x.xx) xxx | xxx (xx.x) | XX.X (XX.X) | XX.X (XX.X) | Normal, n(%) | XX (XX.X) |
| | Median | XXX | XXX | XXX | XX.X | XX.X | Abnormal, n(%) | xx(xx.x) |
| | Min, Max | XXX, XXX | XXX, XXX | XXX, XXX | XX.X, XX.X | XX.X, XX.X | | |
| Day 2, 0.5 hrs | n | XX | XX | XX | XX | XX | | |
| | Mean (SD) | xxx (xx.x) | (x.xx) xxx | xxx (xx.x) | XX.X (XX.X) | XX.X(XX.X) | Normal, n(%) | xx(xx.x) |
| | Median | XXX | XXX | XXX | XX.X | XX.X | Abnormal, n(%) | xx (xx.x) |
| | Min May | ARABAR ARABAR | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | , | , | | | |

Page X of Y

Global Alliance for TB Drug Development Protocol Number: TBI-876-CL-002

Table 14.3.4.2: Summary of 12-Lead ECG Numeric Results
Absolute Values and Change from Baseline by Treatment and Time Point
Safety Population

| | Group 1<br>(N=XX) | Group 2<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| [Tests Name (Units)] | | | |
| Baseline | | | |
| Z | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X(XX.X) | XX.X(XX.X) |
| Median | XX | XX | XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |
| Day 1 Post-Dose [2] | | | |
| Z | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X(XX.X) | XX.X (XX.X) |
| Median | XX | XX | X |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |
| Change from Baseline | | | |
| Z | XX | XX | X |
| Mean (SD) | XX.X (XX.X) | XX.X(XX.X) | XX.X(XX.X) |
| Median | XX | XX | X |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |

# <Continue for all other applicable study days>

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1.

Generated on XX/XX/XX:XXXX by XXX / Uses: XXXX / Reference: Data Listing XXXX

[Programming note: Summarize all ECG tests with continuous results, including ventricular rate, PR, QRS, QT, QTcF intervals. Page break between ECG tests.] Page X of Y

Global Alliance for TB Drug Development Protocol Number: TBI-876-CL-002

Table 14.3.4.3: Summary of 12-Lead ECG Categorical Analysis

Safety Population

| | Group 1<br>(N=XX) | Group 2 $(N=XX)$ | Overall<br>(N=XX) |
|---|---|---|---|
| OTcF (msec) | | | |
| Absolute Values [1] | | | |
| > 450 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| > 480 | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| > 500 | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Change from baseline [2] | | | |
| > 30 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 09 < | XX (XX.X) | XX (XX.X) | XX(XX.X) |

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1.

[1] Subjects with QTcF absolute values > (450, 480 and 500 msec) at any post dosing time point are included. [2] Subjects with QTcF change from baseline values > (30 and 60 msec) at any post dosing time point are included. <a href="#"></a>-Programming Note: Additional QTcF value categories may be added to aid data interpretation.

Generated on XX/XX/XX:XXXX by XXX / Uses: XXXX / Reference: Data Listing XXXX
|<u>E</u> 4

| | sale 17.3.3.1. Summary of Chinear Laboratory 15st results, fromatorings and Coagulation Safety Population | | Safet | Safety Population | <b>.</b> | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | | HCT<br>(ratio) | HGB<br>(g/L) | RBC<br>(10^12/L) | WBC (10^9/L) | PLAT<br>(10^9/L) | RETI<br>(ratio) | aPTT2 (sec) | PT2 (sec) |
| Screening | п | XX | XX | XX | XX | XX | XX | X | XX |
| | Mean (SD) | xxx (xx.x) | xxx (xx.x) | X.XX (X.XX) | x.x(x.x) | XXX (XX.X) | (xxx) xxx. | xx (xx.x) | XX (XX.X) |
| | Median | XXX | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Min, Max | XXX, XXX | XXX, XXX | X.XX, X.XX | X.X, X.X | XXX, XXX | .xxx, .xxx | xx, xx | xx, xx |
| Day -1 | и | XX | XX | XX | XX | X | XX | X | XX |
| | Mean (SD) | XXX (XX.X) | xxx (xx.x) | X.XX (X.XX) | x.x (x.x) | xxx (xx.x) | (xxx.) xxx. | XX (XX.X) | xx (xx.x) |
| | Median | XXX | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Min, Max | XXX, XXX | XXX, XXX | X.XX, X.XX | X.X, X.X | XXX, XXX | .XXX, .XXX | XX, XX | xx, xx |
| Day 2 | и | XX | XX | XX | XX | XX | XX | X | XX |
| | Mean (SD) | XXX (XX.X) | xxx (xx.x) | X.XX (X.XX) | x.x (x.x) | xxx (xx.x) | (xxx.) xxx. | xx (xx.x) | xx (xx.x) |
| | Median | XXX | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Min, Max | XXX, XXX | XXX, XXX | X.XX, X.XX | X.X, X.X | XXX, XXX | .xxx, .xxx | xx, xx | XX, XX |
| | и | XX | XX | XX | XX | XX | XX | XX | XX |
| Day 3 | Mean (SD) | xxx (xx.x) | xxx (xx.x) | x.xx (x.xx) | x.x(x.x) | xxx (xx.x) | (xxx.) xxx. | xx (xx.x) | xx (xx.x) |
| | Median | XXX | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| ote | Min Moy | | | | | | | | |

HCT = Hematocrit; HGB = Hemoglobin; RBC = Erythrocytes; WBC=Leukocytes; PLAT = Platelets, RETI=Reticulocytes, aPTT2=Activated partial thromboplastin time, PT2=Prothrombin time.

| | | NE | NEUT | L | LYM | MO | MONO | E | EOS | BA | BASO |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | | (10^9/L) | 10^9/L) (Ratio) | (10^9/L) | (10^9/L) (Ratio) | (10^9/L) | (10^9/L) (Ratio) | (10^9/L) | (10^9/L) (Ratio) | (10^9/L) | (10^9/L) (Ratio) |
| Screening | п | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | x.x (x.x) | x.xx (x.xx) | x.x (x.x) | $\mathbf{x}.\mathbf{x}\mathbf{x}$ $(\mathbf{x}.\mathbf{x})$ $\mathbf{x}.\mathbf{x}$ $(\mathbf{x}.\mathbf{x})$ $\mathbf{x}.\mathbf{x}$ $(\mathbf{x}.\mathbf{x})$ | x.x (x.x) | x.xx (x.xx) | x.x (x.x) | x.xx (x.xx) | x.x (x.x) | X.XX (X.XX) |
| | Median | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Min, Max | X.X, X.X | X.XX, X.XX | X.X, X.X | X.XX, X.XX | X.X, X.X | X.XX, X.XX | X.X, X.X | X.XX, X.XX | X.X, X.X | X.XX, X.XX |
| Day -1 | п | XX | XX | XX | XX | XX | X | XX | XX | XX | XX |
| | Mean (SD) | x.x (x.x) | x.xx (x.xx) | x.x (x.x) | X.XX(X.XX) $X.X(X.X)$ $X.XX(X.XX)$ $X.X(X.X)$ | x.x (x.x) | x.xx (x.xx) | x.x (x.x) | x.xx (x.xx) | x.x (x.x) | x.xx (x.xx) |
| | Median | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Min, Max | X.X, X.X | X.XX, X.XX | X.X, X.X | X.X, X.X X.XX, X.XX | X.X, X.X | X.XX, X.XX | X.X, X.X | X.X, X.X X.XX, X.XX | X.X, X.X | X.XX, X.XX |
| Day 2 | и | X | XX | XX | XX | XX | X | XX | XX | XX | XX |
| | Mean (SD) | x.x (x.x) | X.XX (X.XX) | x.x (x.x) | $x.xx\left(x.xx\right) x.x\left(x.x\right) x.xx\left(x.x\right) x.x\left(x.x\right) x.xx\left(x.x\right) x.x\left(x.x\right) x.x\left(x.x\right)$ | x.x (x.x) | X.XX (X.XX) | x.x (x.x) | X.XX (X.XX) | x.x (x.x) | x.xx (x.xx) |
| | Median | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Min, Max | X.X, X.X | X.XX, X.XX | X.X, X.X | x.xx, x.xx | X.X, X.X | X.XX, X.XX | X.X, X.X | x.xx, x.xx | X.X, X.X | X.XX, X.XX |
| | и | XX | XX | XX | XX | X | X | XX | XX | XX | XX |
| Day 3 | Mean (SD) | X.X(X.X) | | x.x (x.x) | $x.xx \; (x.xx) x.x \; (x.x) x.x \; (x.xx) x.x $ | x.x (x.x) | x.xx (x.xx) | x.x (x.x) | x.xx (x.xx) | | x.xx (x.xx) |
| | Median | x.x | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| etc | Min May | * * * * | | | | | | | | | |

NEUT = Neutrophils; LYM = Lymphocytes; MONO = Monocytes; EOS = Eosinophils; BASO = Basophils

| TB Alliance |
|---------------------------------|
| Protocol Number: TBAJ-876-CL002 |

Table 14.3.5.3: Summary of Clinical Laboratory Test Results, Electrolytes and Renal Function Safety Population

| | | | Saret | y Population | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | | SODIUM (mmol/L) | K<br>(mmol/L) | CL<br>(mmol/L) | BICARB (mmol/L) | CA<br>(mmol/L) | MG<br>(mmol/L) | UREAN (mmol/L) | CREAT (umol/L) |
| Screening | п | XX | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | XXX (XX.X) | x.x (x.x) | xxx (xx.x) | XX (XX.X) | x.x (x.x) | X.XX (X.XX) | x.x (x.x) | xx (xx.x) |
| | Median | XXX | X.X | XXX | XX | X.X | X.XX | X.X | XX |
| | Min, Max | XXX, XXX | X.X, X.X | XXX, XXX | xx, xx | X.X, X.X | X.XX, X.XX | X.X, X.X | xx, xx |
| Day -1 | п | XX | XX | XX | X | XX | XX | XX | XX |
| | Mean (SD) | XXX (XX.X) | x.x (x.x) | xxx (xx.x) | xx (xx.x) | x.x (x.x) | X.XX (X.XX) | x.x (x.x) | xx (xx.x) |
| | Median | XXX | X.X | XXX | XX | X.X | X.XX | X.X | XX |
| | Min, Max | XXX, XXX | X.X, X.X | XXX, XXX | XX, XX | X.X, X.X | X.XX, X.XX | X.X, X.X | xx, xx |
| Day 2 | п | XX | XX | XX | XX | xx | XX | XX | XX |
| | Mean (SD) | XXX (XX.X) | x.x (x.x) | XXX (XX.X) | XX (XX.X) | x.x (x.x) | X.XX (X.XX) | x.x(x.x) | xx (xx.x) |
| | Median | XXX | X.X | XXX | XX | X.X | X.XX | X.X | XX |
| | Min, Max | XXX, XXX | X.X, X.X | XXX, XXX | XX, XX | X.X, X.X | X.XX, X.XX | X.X, X.X | XX, XX |
| | п | XX | XX | | XX | | XX | XX | XX |
| Day 3 | Mean (SD) | xxx (xx.x) | (x.x)(x.x) | xxx (xx.x) | xx (xx.x) | X.X (X.X) | x.xx (x.xx) | x.x (x.x) | xx (xx.x) |
| | Median | XXX | X.X | | XX | | X.XX | X.X | XX |
| etc | Min, Max | XXX, XXX | X.X, X.X | XXX, XXX | XX, XX | | X.XX, X.XX | X.X, X.X | XX, XX |

K=Potassium, CL=Chloride, BICARB=Bicarbonate, CA=Calcium, MG=Magnesium, UREAN=Urea nitrogen, CREAT=Creatinine

Generated on XX/XX/XX:XXXX by XXXXXX / Uses: XX

[Programming Note: For out of range results, use bold font and superscript L or H]


| | | | Safety Population | oulation | raote 14.5.5.4. Summary of Crimea Laboratory (est Nesuns, Liver runchon) Safety Population | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | | ALT<br>(ukat/L) | AST (ukat/L) | ALP<br>(ukat/L) | TBILI (nmol/L) | DBILI (umol/L) | (umol/L) | LDH<br>(ukat/L) |
| Screening | и | XX | XX | XX | XX | XX | XX | X |
| | Mean (SD) | X.XX(X.XX) | X.XX (X.XX) | (x.xx) xx.x | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.xx (x.xx) |
| | Median | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Min, Max | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX | X.X, X.X | X.X, X.X | X.X, X.X | X.XX, X.XX |
| Day -1 | и | XX | XX | XX | XX | XX | XX | × |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | (xx.x) xx.x | x.x (x.x) | x.x (x.x) | x.x (x.x) | (xx.x) xx.x |
| | Median | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Min, Max | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX | X.X, X.X | X.X, X.X | X.X, X.X | X.XX, X.XX |
| Day 2 | и | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | X.XX (X.XX) | (xx.x) xx.x | x.x (x.x) | x.x (x.x) | x.x (x.x) | (x.xx) |
| | Median | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Min, Max | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX | X.X, X.X | X.X, X.X | X.X, X.X | X.XX, X.XX |
| | п | XX | XX | XX | XX | XX | XX | XX |
| Day 3 | Mean (SD) | x.xx(x.xx) | x.xx (x.xx) | X.XX (X.XX) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.xx(x.xx) |
| | Median | X.XX | X.XX | X.XX | X.X | X.X | X.X | x.xx |
| c to | M. M. | | | | | | | |

ALT=Alanine transaminase, AST=Aspartate transaminase, ALP=Alkaline phosphatase, TBILI=Total bilirubin, DBILI=Direct bilirubin, IBILI=Indirect bilirubin, LDH=Lactate dehydrogenase.


| TB Alliance Protocol Number: TBAJ-876-CL002 | Page 1 of 3 |
|---|---|
| | Table 14.3.5.5: Summary of Clinical Laboratory Test Results, Other Serum Chemistry |
| | Safety Population |

| Time Point | | TPROT<br>(g/L) | GLUC<br>(mmol/L) | ALB<br>(g/L) | URAC<br>(umol/L) | CPK<br>(ukat/L) | AMY<br>(ukat/L) | LIP<br>(ukat/L) |
|---|---|---|---|---|---|---|---|---|
| Screening | и | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | XXX (XX.X) | xx (xx.x) | xxx (xx.x) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Min, Max | xx, xx | XXX, XXX | XX, XX | XXX, XXX | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| Day -1 | п | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | XX (XX.X) | XXX (XX.X) | XX (XX.X) | XXX (XX.X) | X.X | X.XX (X.XX) | x.xx (x.xx) |
| | Median | XX | XXX | XX | XXX | | X.XX | X.XX |
| | Min, Max | XX, XX | XXX, XXX | xx, xx | XXX, XXX | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| Day 2 | п | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | XX (XX.X) | XXX(XX.X) | xx (xx.x) | XXX (XX.X) | X.XX(X.XX) | x.xx (x.xx) | x.xx(x.xx) |
| | Median | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Min, Max | XX, XX | XXX, XXX | XX, XX | XXX, XXX | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| | ٤ | × | × | XX | XX | XX | XX | XX |
| Day 3 | Mean (SD) | XX (XX.X) | XXX (XX.X) | xx (xx.x) | XXX (XX.X) | X.XX (X.XX) | X.XX (X.XX) | X.XX (X.XX) |
| | Median | XX | XXX | X | XXX | x.xx | XX.X | x.xx |
| etc | Min, Max | XX, XX | XXX, XXX | xx, xx | XXX, XXX | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |

TPROT=Total protein, GLUC=Glucose, ALB=Albumin, URAC=Uric acid, CPK=Creatinine phosphokinase, AMY=Amylase, LIP=Lipase


| TB Alliance<br>Protocol Number: | <b>TB Alliance</b><br>Protocol Number: TBAJ-876-CL002 | Table 14. | 4.3.5.6: Summary of Clinical Laboratory Test Results, Urinalysis, Part 1 | linical Laboratory T | est Results. Urinalys | is. Part 1 | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Safety Population | | | | |
| Time Point | | Hd | SpG (g/mL) | GLUC | KET | BILI | CREAT | SOD |
| Screening | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) Abnormai | XX (XX.X) | XX (XX.X) | (x.xx) xx | (x.xx) xx | (X.XX) | (x·xx) xx | xx (xx.x) |
| Day -1 | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) Abnormal | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 2 | n(%) Normal | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) Abnormal | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Day 3 | n(%) Normal | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) Abnormal | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Day 7 | n(%) Normal | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| | n (%) Abnormal | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Day 20 | n(%) Normal | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| | n (%) Abnormal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| etc | | | | | | | | |

SpG=Specific gravity, GLUC=Glucose, KET=Ketones, BILI=Bilirubin, CREAT=Creatinine, SOD=Sodium.

[Programming Note: For out of range results, use bold font and superscript A.]


| | Table | | f Clinical Laboratory<br>Safety Population | 4.3.5.7: Summary of Clinical Laboratory Test Results, Urinalysis, Part 2 Safety Population | iis, Part 2 | |
|---|---|---|---|---|---|---|
| Time Point | | PROT | )<br>) | NIT | LEUK | Microscopic Examination (if indicated) |
| Screening | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | xx (xx.x) |
| | n (%) Abnormal | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| Day -1 | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Day 2 | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| | n (%) Abnormal | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| Day 3 | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| | n (%) Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Day 7 | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Day 20 | n(%) Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) Abnormal | $(x \times x) \times x$ | (x, x, x) | $(x \times x) \times x$ | $(x \times x) \times x$ | (X,XX) |

PROT=Protein, OCC=Occult blood, NIT=Nitrite, LEUK=Leukocyte esterase.

TB Alliance

Protocol Number: TBAJ-876-CL002

Figure 14.2.1: Mean Plasma Midazolam Concentration vs Time Post-dose

PK Population



Note: Concentrations BLOQ are included as 0.

Generated on ... by ... / Uses: ADPC / Reference: Table 14.2.1.2.1.

Note: Use similar formats for all analytes and for individual subject plots.

TB Alliance

Protocol Number: TBAJ-876-CL002

Figure 14.2.3: Mean Plasma Digoxin Concentration vs Time Post-dose

PK Population



Note: Concentrations BLOQ are included as 0.

Generated on ... by ... / Uses: ADPC / Reference: Table 14.2.1.2.1.

TB Alliance

Protocol Number: TBAJ-876-CL002

Figure 14.2.4: Mean Day 17 Plasma TBAJ-876 Concentration vs Time Post-dose





Note: Concentrations BLOQ are included as 0.

Generated on ... by ... / Uses: ADPC / Reference: Table 14.2.1.2.1.

**TB Alliance** Protocol Number: TBAJ-876-CL002

Listing 16.1.7: Subject Enrollment

## All Enrolled Subjects

| ject | Subject Date of Informed Consent | Satisfy All I/E Criteria? | Date-Time of Enrollment | Enrollment Number | Group |
|---|---|---|---|---|---|
| XXX | XX-XX-XXXX | XXX | xxxx-xx-xxTxx:xx | XXX | 1 |
| XXX | XX-XX-XXX | XXX | xxxx-xx-xxTxxxxx | XXX | 1 |
| XXX | XXXXX-XXX | XXX | xxxx-xx-xxTxx:xx | XXX | 1 |

Generated on XX/XX/XX XX:XX by XXXX/ Uses: XXXX

[Programming Note: List all enrolled subjects in order of their date-time of enrollment.]

| TB Alliance Page X | ge X of Y |
|---------------------------------|-----------|
| Protocol Number: TBAJ-876-CL002 | |

Listing 16.2.1.1: Screen Failures

| | Date of | 4 | | | | |
|---|---|---|---|---|---|---|
| Subject | Informed<br>Subject Consent | Date of<br>Screening | Sex | Race | Ethnicity | Reason for Screen Failure |
| XXX | XXXX-XX-XX | XX-XX-XXX | XXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | XX-XX-XXX | XX-XX-XXX | XXXXXXX | XXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | XX-XX-XXX | XX-XX-XXX | XXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | XX-XX-XXX | XX-XX-XXX | XXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | XX-XX-XXX | XX-XX-XXX | XXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | XX-XX-XXX | XX-XX-XXX | XXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | XX-XX-XXX | XX-XX-XXX | XXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX |

Generated on XX/XX/XX:XXXXXXXX by XXXX/ Uses: XXXX

[Programming Note: In Reason for Screen Failure, include list of inclusion criteria not met along with Primary Reason for Screen Failure and Comments (IECOMM).]

| | | Completion Status |
|---|---|---|
| | Disposition ects | Date of Last Contact Completion Status |
| | Listing 16.2.1.2: Subject Disposition<br>All Enrolled Subjects | Date of Last Visit |
| | | Date Enrolled |
| B Alliance<br>rotocol Number: TBAJ-876-CL002 | | Screening Date |
| TB Alliance<br>Protocol Number | | Subject |

XXXXXXXXXXXXXXXXX

XXXXXXXXXXXXXXXXXXX

(XX) XX-XX-XXX XXX XXX XX-XX-XXX (XX) XX-XX-XXX XXX

(xx) xx-xx-xxx

XXXX-XX-XX (1) XXXX-XX-XX (1) XXXX-XX-XX (1)

(XX-) XXX-XX-XXX (-XX) XXXX-XX-XX (-XX) XXXX-XX-XX (-XX) XXXX-XX-XX (-XX) XXX-XX-XX-XX (-XX) XXX-XX-XX-XX-XX

\* \* \* \* \* \*

XXX

(xx) xx-xx-xxx (xx) xx-xx-xxxx

(XX) XX-XX-XXXX

xxxx-xx-(1)

xxx-xx-xx(1)xxxx-xx-xx(1)

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

[Programming Note: Study completion status will include reason for discontinuation (DSDECOD and DSCMTS)]


| Protocol Nun | Protocol Number: TBAJ-876-CL002 | 76-CL002 | | | 1 486 A 01 1 |
|---|---|---|---|---|---|
| | | | Listing 16.2.2: I<br>All Enrol | Listing 16.2.2: Protocol Deviations<br>All Enrolled Subjects | |
| Subject | Subject Category | Date (Day) | Protocol Deviation | Protocol Deviation Type | Action Taken |
| XXX | Major<br>Major | (x) xx-xx-xxxx (x) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | Major | (XX) XX-XX-XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TB Alliance
Protocol Number: TBAJ-876-CL002

Listing 16.2.4.1: Demographics and Baseline Characteristics All Enrolled Subjects

| | | | , a | 77 | Weight (kg) | (kg) | | |
|---|---|---|---|---|---|---|---|---|
| Subject | ubject Age | Gender <sup>R</sup> | Kace | Ethnicity | Screening Day -1 | Day -1 | Height (cm) BMI (kg/m²) | $BMI (kg/m^2)$ |
| XXX | XX | Male | XXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX.X | XX.X | XXXX.X | XX.X |
| XXX | XX | Female | XXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX.X | XX.X | XXXX.X | XX.X |
| XXX | XX | Male | XXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX.X | XX.X | XXX.X | XX.XX |
| XXX | XX | Female | XXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX.X | XX.X | XXX.X | XX.X |
| XXX | XX | Female | XXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX.X | XX.X | XXX.X | XX.X |
| XXX | XX | Male | XXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX.X | XX.X | XXX.X | XX.X |

Note: BMI = Body Mass Index


| TB Alliance Protocol Nun | TB Alliance<br>Protocol Number: TBAJ-876-CL002 | L002 | | Page X of Y |
|---|---|---|---|---|
| | | Listing 16.2.4.2: Pri | Listing 16.2.4.2: Prior and Concomitant Medication Safety Population | |
| Subject | Prior or<br>Concomitant? | WHO Preferred Term (Verbatim Term) / ATC Classification | Indication /<br>Dose Unit / Frequency / Route | Start Date (Day)-Stop Date (Day) |
| XXX | Concomitant | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | - (xx) xx-xx-xxxx (xx) - (xx) x-xx-xxxxx |
| Note: Study | day is shown only i | Note: Study day is shown only if it is on or after Day 1, or within 30 days prior to Day 1 | ay 1. | |

[Programming Note: List medications in ascending order of start date for each subject.]


| TB Alliance Protocol Nun | TB Alliance Protocol Number: TBAJ-876-CL002 | | | Page X of Y |
|---|---|---|---|---|
| | | Listing 16.2.4.3: Medical History<br>Safety Population | | |
| Subject | Subject Diagnosis | Start Date (Day) | End Date (Day) | Medication Taken Currently? |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (xx) xx-xx-xxxx | (xx) xx-xx-xxxx | XXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (XX) XX-XX-XXX | Ongoing | XXX |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (xx) xx-xx-xxxx | (xx) xx-xx-xxxx | XXX |
| Note: Study of | Note: Study day is shown only if it is within 30 days prior to Day 1. | | | |


| | | | Lis | sting 16.2. | 5.1: Plasm<br>PK I | Listing 16.2.5.1: Plasma Midazolam Concentrations PK Population | am Concer | ıtrations | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Day | Day | Date-time of<br>Dosing | | Pre-<br>dose | 15<br>mins | 30<br>mins | 1 hr | 2 hrs | 3 hrs | 4 hrs | 6 hrs | 8 hrs | 12 hrs | 24 hrs |
| XXX | - | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX:XX |
| | 20 | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX:XX | XX:XX | XX:XX<br>XX:XX |
| XXX | - | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX:XX | XX:XX<br>XX.XX | XX:XX |
| | 20 | xxxx-xx-xxTxx:xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX |


| | | | Listing | 16.2.5.2: F | lasma 1-H<br>PK F | Listing 16.2.5.2: Plasma 1-Hydroxymidazolam Concentrations PK Population | lazolam C | oncentratic | suc | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Day | Day | Date-time of<br>Dosing | | Pre-<br>dose | 15<br>mins | 30<br>mins | 1 hr | 2 hrs | 3 hrs | 4 hrs | 6 hrs | 8 hrs | 12 hrs | 24 hrs |
| XXX | - | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX<br>XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX:XX |
| | 20 | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| XXX | П | xxxx-xx-xxTxx:xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | 20 | xxxx-xx-xxTxx:xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX |


| I <b>5 Alliance</b><br>Protocol Nur | ance<br>I Numbe | IB Alliance<br>Protocol Number: TBAJ-876-CL002 | | Listing 1 | 6.2.5.3: ] | Plasma Digoxi<br>PK Population | Listing 16.2.5.3: Plasma Digoxin Concentrations PK Population | oncentra | tions | | | | | | Fage | rage A of Y |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subj | Day | Date-time of<br>Dosing | | Pre-<br>dose | 30<br>mins | 1 hr | 1 hr 2 hrs 3 hrs | 3 hrs | 4 hrs | 6 hrs | 8 hrs | 12<br>hrs | 24<br>hrs | 48<br>hrs | 72<br>hrs | 96<br>hrs |
| XXX | 2 | xxxx-xx-xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX |
| | 21 | xxxx-xx-xxTxx:xx Sample Time<br>Concentration | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX |
| XXX | 7 | xxxx-xx-xxTxx:xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX |
| | 21 | xxxx-xx-xxTxx:xx Sample Time<br>Concentration | Sample Time xx.xx<br>Concentration (ng/mL) xx.xx | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX |


| | | | Li | sting 16.2 | 5.4: Plas<br>PK | lasma TBAJ-8'<br>PK Population | -876 Con | Listing 16.2.5.4: Plasma TBAJ-876 Concentrations PK Population | S. | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Day | Date-time of<br>Dosing | | Pre-<br>dose | 30<br>mins | 3 hrs | 4 hrs | 5 hrs | 6 hrs | 7 hrs | 8 hrs | 12 hrs | 12 hrs 16 hrs | 20 hrs | 24<br>hrs |
| XXX | 17 | xxxxxxxxxxxxxxx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX:XX | XX:XX | XX:XX | XX:XX |
| xxx | 17 | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX<br>XX.XX |
| xxx | 17 | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX |
| xxx | 17 | xxxx-xx-xxxx | Sample Time<br>Concentration (ng/mL) | XX:XX<br>XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX:XX | XX:XX | XX:XX | XX:XX |


| TB Alliance Protocol Nur | nce<br>Number | TB Alliance Protocol Number: TBAJ-876-CL002 | | | | | | | | | | | | Page | Page X of Y |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Listing | 16.2.5.5: I<br>PK | 5: Plasma M2 (<br>PK Population | Listing 16.2.5.5: Plasma M2 Concentrations PK Population | trations | | | | | | | |
| Subject Day | Day | Date-time of<br>Dosing | | Pre-<br>dose | 30<br>mins | 3 hrs | 4 hrs | 5 hrs | 6 hrs | 7 hrs | 8 hrs | 12 hrs | 12 hrs 16 hrs | 20 hrs | 24<br>hrs |
| XXX | 17 | xx:xxTxx-xx-xxx | Sample Time<br>Concentration (ng/mL) | XX.XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| XXX | 17 | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX |
| XXX | 17 | xx:xxTxx-xx-xxx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX:XX |
| XXX | 17 | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX.XX |


| TB Alliance Protocol Nur | nce<br>Number | TB Alliance Protocol Number: TBAJ-876-CL002 | | | | | | | | | | | | Page | Page X of Y |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Listing | 16.2.5.6: I<br>PK | 5: Plasma M3 (<br>PK Population | Listing 16.2.5.6: Plasma M3 Concentrations PK Population | trations | | | | | | | |
| Subject Day | Day | Date-time of<br>Dosing | | Pre-<br>dose | 30<br>mins | 3 hrs | 4 hrs | 5 hrs | 6 hrs | 7 hrs | 8 hrs | 12 hrs | 12 hrs 16 hrs | 20 hrs | 24<br>hrs |
| XXX | 17 | xx:xxTxx-xx-xxx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX:XX |
| XXX | 17 | xxxx-xx-xxTxx:xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX:XX |
| XXX | 17 | xx:xxTxx-xx-xxx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX:XX | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX:XX | XX:XX<br>XX:XX |
| XXX | 17 | xxxx-xx-xxTxx.xx | Sample Time<br>Concentration (ng/mL) | XX:XX | XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX:XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX<br>XX.XX | XX:XX | XX:XX<br>XX.XX |


| Ocol Nimber: TBA I-876-CI 002 |
|-------------------------------|

| | | | AUC <sub>0-last</sub> | AUC <sub>0-inf</sub> | Cmax | tmax | Kei | t1/2 | CL/F | Vz/F |
|---|---|---|---|---|---|---|---|---|---|---|
| Subj | Day | Day Date-time of Dosing (ng.hr/mI | (ng.hr/mL) | (ng.hr/mL) | (ng/mL) | (hr) | (/hr) | (hr) | (L/hr) | (L) |
| XXX | | xxxxx-xx-xxxxx | XXXX | XXXX | XX.X | X.XX | X.XXXX | X.X.X | XX.X | X.XX |
| | 20 | xx:xxTxx-xx-xxx | XXXX | XXXX | XX.X | x.xx | X.XXXX | X.X.X | XX.X | X.X.X |
| XXX | _ | xx:xxTxx-xx-xxx | XXXX | XXXX | XX.X | X.XX | X.XXXX | X.XX | XX.X | XX.X |
| | 20 | xx:xxTxx-xx-xxx | XXXX | XXXX | XX.X | X.XX | X.XXXX | X.XX | XX.X | XX.X |
| XXX | _ | xxxx-xx-xxTxx:xx | XXXX | XXXX | XX.X | X.XX | X.XXXX | X.XX | XX.X | XX.X |
| | 20 | xxxx-xx-xxTxx:xx | XXXX | XXXX | XX.X | X.XX | X.XXXX | X.XX | XX.X | XX.X |


| TB Alliance Protocol Num | e<br>mber: TBAJ | TB Alliance Protocol Number: TBAJ-876-CL002 | | | | | | | | Page X of Y |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Listing 16.2 | Listing 16.2.6.2: 1-Hydroxymidazolam Pharmacokinetic Parameters PK Population | ymidazolam Pharm<br>PK Population | nacokinetic Pan | ameters | | | |
| Subj | Day | Date-time of Dosing | AUC <sub>0-last</sub> (ng.hr/mL) | AUC <sub>0-inf</sub> (ng.hr/mL) | C <sub>max</sub> (ng/mL) | t <sub>max</sub> (hr) | kei<br>(/hr) | t <sub>1/2</sub> (hr) | CL/F<br>(L/hr) | Vz/F<br>(L) |
| XXX | 1 20 | xxxx-xx-xxTxx:xx<br>xxxx-xx-xxTxx:xx | XXXX | XXXX | XXX.X<br>XXX.X | X.XX<br>X.XX | X.XXXX<br>X.XXXX | X.XX<br>X.X | XX.X<br>XX.X | XX.X<br>XX.X |
| XXX | 1 20 | xxxx-xx-xxTxx.xx<br>xxxx-xx-xxTxx.xx | XXXX | XXXX | XXXX<br>XXXX | X.XX<br>X.XX | X.XXXX<br>X.XXXX | X. XX<br>X. X. | XX.X<br>XX.X | XXX<br>XXXX |
| XXX | 1 20 | XXXXX-XX-XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX | XXXX | XX.X<br>XX.X | X.XX<br>X.XX | X.XXXX<br>X.XXXX | XX.X<br>X.XX | XX.X<br>XX.X | XX.X<br>XX.X |


| Number: TBAJ-876-CL002 | | | | Listi | ing 16.2.6.3: Digc<br>Pl | oxin Pharmacoki<br>K Population | netic Paramete | S | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX-XX-XX-XXXXX XXXX XXXX XXXX XXXX XXXX XXXX-XX-XX-XX-XX-XX-XX-XX-XXXX XXXX XXXXX XXXX XXXX XXXX < | Subj | Day | Date-time of Dosing | AUC <sub>0-last</sub> (ng.hr/mL) | AUC <sub>0-inf</sub> (ng.hr/mL) | C <sub>max</sub> (ng/mL) | t <sub>max</sub> (hr) | kel<br>(/hr) | t <sub>1/2</sub> (hr) | CL/F<br>(L/hr) | Vz/F<br>(L) |
| 2 xxxx-xx-xx-xxTxx.xx xxxx xxxx xxxx xxxx xxxx 21 xxxx-xx-xx-xxTxx.xx xxxx xxxx xxxx xxxx xxxx 2 xxxx-xx-xx-xxTxx.xx xxxx xxxx xxxx xxxx xxxx 21 xxxx-xx-xx-xxTxx.xx xxxx xxxx xxxx xxxx | XXX | 2 21 | xx:xxTxx-xx-xxxx | XXXX | XXXX | XX.X<br>XX.X | X.XX<br>X.XX | X.XXXX<br>X.XXXX | XXX<br>XXXX | XX.X<br>XX.X | XX.X<br>XX.X |
| 2 xxxx-xx-xx-xxTxx.xx xxxx xxxx xx.x x.xx x.x | XXX | 2 21 | XXXX-XX-XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX | XXXX | X.X.X | X.XX<br>X.XX | X.XXXX<br>X.XXXX | XX.X<br>XX.X | XX.X | XX.X<br>XX.X |
| | XXX | 2 21 | XXXX-XX-XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX | XXXX | X.X. | XX.X<br>XXX. | X.XXXX<br>X.XXXX | XXX<br>XXX | XX.X<br>XX.X | XXXX<br>XXXX |

TB Alliance
Protocol Number: TBAJ-876-CL002

| | | 4 | xx | xx | xx | xx | xx | XX | xx |
|---|---|---|---|---|---|---|---|---|---|
| | | 24 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 23 | XX:XX | xx:xx | XX:XX | xx:xx | XX:XX | XX:XX | xx:xx |
| | | 22 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 21 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 20 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 19 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 18 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 17 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| 5 Dosing<br>ts | (Day) | 16 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| BAJ-876<br>d Subject | Time of Dosing (Day) | 15 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | xx:xx | XX:XX |
| Listing 16.2.6.4: TBAJ-876 Dosing<br>All Enrolled Subjects | Time o | 14 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | xx:xx | XX:XX |
| Listing 1<br>A | | 13 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 12 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 11 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 10 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 6 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 8 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 7 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | 9 | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX | XX:XX |
| | | Subj | XXX | XXX | XXX | XXX | XXX | XXX | XXX |


| TB Alliance Protocol Number: TBAI-876-CL002 | Page X of Y |
|---|---|
| Listing 16.2.6.5: TBAJ-876 Day 17 Pharmacokinetic Parameters PK Population | |

| | | TBAJ-876 | 92 | | | M2 | | | | M3 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | AUC <sub>0-24</sub><br>Subj (ng.hr/mL) | C <sub>max</sub> (ng/mL) | t <sub>max</sub> (hr) | Ctrough (ng/mL) | AUC <sub>0-24</sub> (ng.hr/mL) | C <sub>max</sub> (ng/mL) | t <sub>max</sub> (hr) | Ctrough (ng/mL) | AUC <sub>0-24</sub> (ng.hr/mL) | C <sub>max</sub> (ng/mL) | t <sub>max</sub> (hr) | Ctrough (ng/mL) |
| , | | | | | | | | | | | | |
| XXX | XXXX | XX.X | X.XX | XX.X | XXXX | XX.X | X.XX | X.XX | XXXX | XX.X | XX.X | XX.X |
| XXX | XXXX | XX.X | X.XX | X.X.X | XXXX | XX.X | X.XX | X.XX | XXXX | XX.X | XX.X | XX.X |
| × | XXXX | XXX.X | X.XX | X.X.X | XXXX | XX.X | X.XX | X.XX | XXXX | XX.X | X.XX | XX.X |
| × | XXXX | XXX.X | X.XX | X.X.X | XXXX | XX.X | X.XX | X.XX | XXXX | XX.X | X.XX | XX.X |
| × | XXXX | XX.X | X.XX | X.X.X | XXXX | XX.X | X.XX | X.XX | XXXX | XX.X | XX.X | XX.X |
| XXX | XXXX | XX.X | X.XX | X.X.X | XXXX | XX.X | X.XX | X.XX | XXXX | XX.X | XX.X | XX.X |
| × | XXXX | XX.X | X.XX | X.X.X | XXXX | XX.X | X.XX | X.XX | XXXX | XX.X | XX.X | XX.X |
| × | XXXX | XX.X | X.XX | XX.X | XXXX | XX.X | X.XX | X.X.X | XXXX | XX.X | X.XX | XX.X |

TB Alliance
Protocol Number: TBAJ-876-CL002

Listing 16.2.7.1: Adverse Events Safety Population

| Med] (Ver] Med] | MedDRA Preferred Term<br>(Verbatim Term) /<br>Subject MedDRA SOC Term | Start Date-Time (Day) - Stop Date-Time (Day) / Date-Time (Day) Reported | TEAE? / Severity / Outcome / Relationship to Study Drug (Regimen*) | Action Taken with Study Product /<br>Other Action Taken /<br>Serious? (Criteria Met) |
|---|---|---|---|---|
| XXXXXXX<br>XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx.xx (xx) – xxxx-xx-xxTxx.xx (xx) / xxxx-xx-xxTxx.xx (xx) | xxx / xxxxxxxx / xxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXX / XXXXXXXXXXX / XXXXXXXX |
| XXXXXXX<br>(XXXXXXX) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx:xx (xx) – Ongoing / xxxx-xx-xxTxx:xx (xx) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx.xx (xx) – xxxx-xx-xxTxx.xx (xx) / xxxx-xx-xxTxx.xx (xx) | xxx / xxxxxxxx / xxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXXX / XXXXXXXXXXXXXXXX / XX |

TEAE= Treatment-emergent adverse event (onset on or after Day 1); SOC=System organ class

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX

\*Note: For Relationship to Study Drug Regimen, show "Not related" if data show "Not related" for all study products. Otherwise, list degree of relationship and attributed regimen (TBAJ-876, midazolam, digoxin, TBAJ-876 plus midazolam, etc).

TB Alliance
Protocol Number: TBAJ-876-CL002

Listing 16.2.7.2: Serious Adverse Events and Adverse Events Leading to Study Discontinuation Safety Population

| <br>MedDRA Preferred Term<br>(Verbatim Term) /<br>Subject MedDRA SOC Term | Start Date-Time (Day) -<br>Stop Date-Time (Day) /<br>Date-Time (Day) Reported | TEAE? / Severity / Outcome / Relationship to Study Drug Regimen | Action Taken with Study Product /<br>Other Action Taken /<br>Serious? (Criteria Met) |
|---|---|---|---|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx:xx (xx) -<br>xxxx-xx-xxTxx:xx (xx) /<br>xxxx-xx-xxTxx:xx (xx) | XXXXXXXXX / XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xx1xx:xx (xx) – Ongoing / xxxx-xx-xxTxx:xx (xx) | XXXXXXXXX / XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXX / XXXXXXXXXXXXXXXXXX / XX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx:xx (xx) – xxxx-xx-xxTxx:xx (xx) / xxxx-xx-xxTxx:xx (xx) | / xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXXX / XXXXXXXXXXXX / XXXXXX |

TEAE= Treatment-emergent adverse event (onset on or after Day 1); SOC=System organ class

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX

Note: For Relationship to Study Drug Regimen, show "Not related" if data show "Not related" for all study products. Otherwise, list degree of relationship and attributed regimen (TBAJ-876, midazolam, digoxin, TBAJ-876 plus midazolam, etc).

Protocol Number: TBAJ-876-CL002 TB Alliance

Listing 16.2.7.3: Cardiovascular Adverse Events Safety Population

| | | | Saicty i opalation | | |
|---|---|---|---|---|---|
| Subject | MedDRA Preferred Term<br>(Verbatim Term) /<br>Subject MedDRA SOC Term | Start Date-Time (Day) -<br>Stop Date-Time (Day) /<br>Date-Time (Day) Reported | TEAE? / Severity / Outcome / Relationship to Study Drug Regimen | Action Taken with Study<br>Product /<br>Other Action Taken /<br>Serious? (Criteria Met) | Vital Signs Taken Closest to<br>Cardiovascular Event:<br>Systolic BP (mmHg)/Diastolic<br>BP (mmHg) (Heart Rate<br>(bpm)) |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx:xx (xx) – xxxx-xx-xxTxx:xx (xx) / xxxx-xx-xxTxx:xx (xx) | XXX / XXXXXXXXX / XXXXXXXXXXXX / XXXXXXX | XXXXXXXXXXXXXXXX / XXXXXXXXXXXXXXXXXXX | xx/xx (xx) |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx:xx (xx) – Ongoing / xxxx-xx-xxTxx:xx (xx) | XXX / XXXXXXX / XXXXXXXX / XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxx/xx (xx) |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx:xx (xx) –<br>xxxx-xx-xxTxx:xx (xx) /<br>xxxx-xx-xxTxx:xx (xx) | xxx /<br>xxxxxxxx /<br>xxxxxxxxxxxxxxx / | XXXXXXXXXXXXXXX / XXXXXXXXXXXXXXXXXXXXX | xxx/xx (xx) |

TEAE= Treatment-emergent adverse event (onset on or after Day 1); SOC=System organ class

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

Note: For Relationship to Study Drug Regimen, show "Not related" if data show "Not related" for all study products. Otherwise, list degree of relationship and attributed regimen (TBAJ-876, midazolam, digoxin, TBAJ-876 plus midazolam, etc).

TB Alliance Protocol No. TBAJ-876-CL002 TKL No. P1980322 Page X of Y Presence of Heart Murmur XXX XXX XXX XXX XXX XXX XXX  $\mathbf{X}\mathbf{X}\mathbf{X}$  $\mathbf{X}\mathbf{X}\mathbf{X}$ Listing 16.2.8.1: Physical Examinations Safety Population Findings Normal Normal Normal Normal Normal Normal Normal XXXXXXXXXXX XXXXXXXXXXX **Body System** All systems All systems All systems All systems All systems All systems All systems (x-) xx:xxTxx-xx-xxxx (x-) xx:xxTxx-xx-xxxx (x-) xx:xxTxx-xx-xxxx (x) xx:xxTxx-xx-xxx (x) xx:xxTxx-xx-xxx (x) xx:xxTxx-xx-xxx (x) xx:xxTxx-xx-xxx(x) xx:xxTxx-xx-xxx Date-Time (Day) Protocol Number: TBAJ-876-CL002 Time Point Day 25/ET Screening Screening Day -1 Day 5 Day 2 Day 3 Day 4 Subject TB Alliance XXX XXX

Note: Full physical examination includes HEENT, neck, heart, respiratory, abdomen, musculoskeletal, neurological status, skin, and other. Body systems were normal if not otherwise shown.

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

etc


| | | | | | Sarety Population | tion | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subj | Time Point | Time Point Date-Time (Day) | Supine<br>Systolic<br>BP<br>(mmHg) | Supine<br>Diastolic<br>BP<br>(mmHg) | Supine<br>Heart<br>Rate<br>(bpm) | Temp<br>(C) | Resp Rate (bpm) | Pulse<br>Oximetry<br>(%) | Supine<br>Systolic<br>BP<br>(mmHg) | Supine<br>Diastolic<br>BP<br>(mmHg) | Supine<br>Heart<br>Rate<br>(bpm) |
| | | F | | | | | | | | | |
| XXX | Screening | (x-) xx:xx1xx-xx-xxx | XXX | XXX | XXX | X.XX | XX | X.XX | XXX | XXX | XXX |
| | Day -1 | (x-) xx:xxTxx-xx-xxx | XXX | XXX | XXX | XX.X | X | X.X.X | XXX | XXX | XXX |
| | Day 1 | (x-) xx:xxTxx-xx-xxxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Pre-dose | xxxx-xx-xxTxx:xx(x) | xxx | xxx | xxx | XX.X | XX | XXX.X | xxx | xxx | XXX |
| | 0.5 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | xxx | X.X.X | xx | XXX.X | xxx | xxx | XXX |
| | 1 hr | xxxx-xx-xxTxx:xx(x) | XXX | XXX | xxx | X.X.X | xx | XXX.X | xxx | XXX | XXX |
| | 2 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 6 hrs | xxxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | X.X.X | xx | XX.X | XXX | XXX | XXX |
| | 12 hrs | xxxxx-xx-xxTxx | XXX | XXX | xxx | X.X.X | xx | XX.X | xxx | XXX | XXX |
| | Day 2 | xxxxx-xx-xxTxx | XXX | XXX | XXX | X.XX | XX | XX.X | XXX | XXX | XXX |
| | Pre-dose | xxxxx-xx-xxTxx | XXX | XXX | xxx | X.X.X | xx | XX.X | xxx | XXX | XXX |
| | 0.5 hrs | xxxxx-xx-xxTxx | XXX | XXX | xxx | X.X.X | xx | XX.X | xxx | xxx | XXX |
| | 1 hr | xxxxx-xx-xxTxx | XXX | XXX | xxx | X.X.X | xx | XX.X | xxx | XXX | XXX |
| | 2 hrs | xxxxx-xx-xxTxx | XXX | XXX | xxx | X.X.X | xx | XX.X | xxx | XXX | XXX |
| | 6 hrs | xxxxx-xx-xxTxx | XXX | XXX | xxx | X.X.X | xx | XX.X | xxx | XXX | XXX |
| | 12 hrs | xxxxx-xx-xxTxx | XXX | XXX | xxx | X.X.X | xx | XX.X | xxx | XXX | XXX |
| | Day 6 | xxxxx-xx-xxTxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Pre-dose | xxxx-xx-xxTxx:xx(x) | XXX | XXX | xxx | X.X.X | xx | XXX.X | xxx | XXX | XXX |
| | 0.5 hrs | xxxxx-xx-xxTxx | xxx | XXX | xxx | x.xx | xx | XX.X | xxx | xxx | XXX |
| | 1 4 1 | (a) and the Tark that the territories | ***** | , | | ** *** | , | | | , | 444 |
| | III | | YYY | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | VVV |

Note: On Days 7 through 19, vital signs are taken 6 hours after dosing. Supine measurements are taken after at least 2 minutes in supine position, and standing measurements are taken after at least 1 minute standing.


| | | | | | salety Population | tion | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subj | Time Point | Date-Time (Day) | Supine<br>Systolic<br>BP<br>(mmHg) | Supine<br>Diastolic<br>BP<br>(mmHg) | Supine<br>Heart<br>Rate<br>(bpm) | Temp<br>(C) | Resp Rate<br>(bpm) | Pulse<br>Oximetry<br>(%) | Supine<br>Systolic<br>BP<br>(mmHg) | Supine<br>Diastolic<br>BP<br>(mmHg) | Supine<br>Heart<br>Rate<br>(bpm) |
| XXX | Day 6 | xxxx-xx-xxTxx:xx (-x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 6 hrs | (x-) xx::xxTxx-xx-xxx | XXX | XXX | XXX | X.X.X | XX | XX.X | XXX | XXX | XXX |
| | 12 hrs | (x-) xx:xxTxx-xx-xxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 7 | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 8 | xxxx-xx-xxTxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 9 | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 10 | xxxx-xx-xxTxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 11 | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | xx.x | XXX | XXX | XXX |
| | Day 12 | xxxxx-xx-xx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 13 | XXXX-XX-XXTXX:XX(X) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 14 | xxxxx-xx-xx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 15 | XXXX-XX-XXTXX:XX(X) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 16 | xxxxxxxxxxxxxxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 17 | xxxxxxxxxxxxxxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 18 | xxxxxxxxxxxxxxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 19 | xxxxxxxxxxxxxxxxxxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 20 | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Pre-dose | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 0.5 hrs | xxxxxxxxxxxxxxxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 1 hr | xxxxx-xx-xxTxx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |

Note: On Days 7 through 19, vital signs are taken 6 hours after dosing. Supine measurements are taken after at least 2 minutes in supine position, and standing measurements are taken after at least 1 minute standing.


| TB Alliance Protocol Nun | TB Alliance<br>Protocol Number: TBAJ-876-CL002 | 1-876-CL002 | | | | | | | | d | Page X of Y |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Listing 16.2. | Listing 16.2.8.2: Vital Signs Measurements<br>Safety Population | s Measureme<br>ion | nts | | | | |
| Subj | Time Point | Date-Time (Day) | Supine<br>Systolic<br>BP<br>(mmHg) | Supine<br>Diastolic<br>BP<br>(mmHg) | Supine<br>Heart<br>Rate<br>(bpm) | Temp<br>(C) | Resp Rate<br>(bpm) | Pulse<br>Oximetry<br>(%) | Supine<br>Systolic<br>BP<br>(mmHg) | Supine<br>Diastolic<br>BP<br>(mmHg) | Supine<br>Heart<br>Rate<br>(bpm) |
| XXX | Day 20 | xxxx-xx-xxTxx:xx (-x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 6 hrs | | XXX | xxx | xxx | XX.X | xx | XX.X | XXX | xxx | XXX |
| | 12 hrs | xxxx-xx-xxTxx.xx | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Day 21 | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | Pre-dose | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 0.5 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 1 hr | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |
| | 2 hrs | xxxx-xx-xxTxx:xx(x) | XXX | xxx | XXX | XX.X | xx | x.xx | XXX | XXX | XXX |
| | 6 hrs | xxxx-xx-xxTxx:xx(x) | xxx | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | xxx |
| | 12 hrs | xxxx-xx-xxTxx:xx(x) | xxx | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | xxx |
| | Day 24 | xxxx-xx-xxTxx:xx(x) | xxx | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | xxx |
| | Pre-dose | xxxx-xx-xxTxx:xx(x) | xxx | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | xxx |
| | 0.5 hrs | xxxx-xx-xxTxx:xx(x) | xxx | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | xxx |
| | 1 hr | XXXX-XX-XXXXXX | XXX | xxx | XXX | XX.X | xx | x.xx | XXX | XXX | xxx |
| | 2 hrs | xxxx-xx-xxTxx:xx(x) | xxx | xxx | xxx | XX.X | xx | XX.X | xxx | xxx | xxx |
| | 6 hrs | xxxx-xx-xxTxx:xx(x) | xxx | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | xxx |
| | 12 hrs | xxxx-xx-xxTxx:xx(x) | xxx | xxx | XXX | XX.X | XX | XX.X | XXX | XXX | xxx |
| | Day 25/ET | xxxx-xx-xxTxx:xx (x) | XXX | XXX | XXX | XX.X | XX | XX.X | XXX | XXX | XXX |

Note: On Days 7 through 19, vital signs are taken 6 hours after dosing. Supine measurements are taken after at least 2 minutes in supine position, and standing measurements are taken after at least 1 minute standing.


| | | | | Sal | Safety Population | Lisung 10.2.8.3: Electrocardiogram (ECG) Resuits<br>Safety Population | 3 | |
|---|---|---|---|---|---|---|---|---|
| Subject | Time Point | Date-Time (Dav) | HR<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF<br>(msec) | Investigator's Assessment / Comments |
| | 2 31 35 35 5 | (*) *********************************** | | | | | | |
| XXX | Scieening<br>Dav -1 | (x-) xx.xx1xx-xx-xxxx (x-) | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX | XXX | *************************************** |
| | Day 2 | (x-) xx:xxTxx-xx-xxxx | XXX | XXX | XXX | XXX | XX | XXXXXXXXXXXXXX |
| | Pre-dose | xxxx-xx-xxTxx:xx (x) | XXX | XXX | xxx | xxx | XXX | XXXXXXXXXXXXXXXXXX |
| | 0.5 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXX |
| | 1 hr | xxxxx-xx-xxTxx:xx (x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXX |
| | 2 hrs | xxxxx-xx-xxTxx | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXX |
| | 6 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | 12 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | Day 3 | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | Day 7 | xxxxx-xx-xxTxx | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXX |
| | Day 20 | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | Day 21 | xxxx-xx-xxTxx | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXX |
| | Pre-dose | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | 0.5 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | 1 hr | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | 2 hrs | xxxxx-xx-xxTxx | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXX |
| | 6 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | 12 hrs | xxxx-xx-xxTxx:xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXX |
| | Day 22 | xxxx-xx-xxTxx.xx(x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXXXXXX |
| | Day 25/ET | xxxx-xx-xxTxx:xx (-x) | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXXXXXXX |

HR=Heart rate, PR=PR interval, QRS=QRS duration, QT=QT interval, QTcF=Corrected QT interval; ET=Early termination.

Generated on XX/XX/XX:XXXX by XXXXXX / Uses: XX

Note: Blank line after every subject. Repeat subject number at the top of each page.


| TB Alliance | | | | | | Page X of Y |
|---|---|---|---|---|---|---|
| Protocol Number: TBAJ-876-CL002 | | | | | | ) |
| | Listing 16.2.8.4.1: Cli | 5.2.8.4.1: Clinical Laboratory Test Results, Hematology and Coagulation | Test Results, Ho | ematology and | Coagulation | |
| | | Safety | Safety Population | | | |
| | | 4011 | Cad | Carr | E + 100 | 6 |

| | | | | Safet | Satety Population | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Subject Time Point | Date-Time (Day) | HCT<br>(ratio) | HGB<br>(g/L) | RBC<br>(10^12/L) | WBC (10^9/L) | PLAT (10^9/L) | RETI<br>(ratio) | aPTT2<br>(sec) | PT2 (sec) |
| | | E | | | | | | | | |
| XXX | Screening | (x-)xx.xx.xx.xx.xx | XXX. | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Day -1 | xxx-xx-xxTxx | XXX. | xxx | X.XX | X.X | xxx | XXX. | xx | XX |
| | Day 2 | xxxx-xx-xxTxxx.xx(x) | XXX. | XXX | X.XX | x.x | XXX | XXX. | XX | XX |
| | Day 3 | xxxx-xx-xxTxxx.xx(x) | .xxx L | XXX | X.XX | x.x | XXX | XXX. | XX | XX |
| | Day 7 | xxxx-xx-xxTxxxxx(x) | XXX. | XXX | X.XX | x.x | XXX | XXX. | XX | XX |
| | Day 20 | xxx-xx-xxTxx:xx(xx) | XXX. | XXX | X.XX | x.x | XXX | XXX. | XX | XX |
| | Day 21 | xxxx-xx-xxTxx:xx (xx) | .xxx L | XXX | X.XX | x.x | XXX | XXX. | XX | XX |
| | Day 22 | xxx-xx-xxTxx | .XXX L | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Day 25/ET | xxxx-xx-xxTxx:xx (xx) | XXX. | XXX | X.XX | X.X | xxx | XXX. | xx | XX |
| XXX | Screening | (x-) $XX:XXTXX-XX-XXX$ | XXX. | XXX | X.XX | x.x | xxx | XXX. | XX | xx |
| | Day -1 | xxx-xx-xxTxx:xx | XXX. | xxx | X.XX | x.x | xxx | XXX. | XX | xx |
| | Day 2 | xxxx-xx-xxTxxxxx(x) | XXX. | xxx | X.XX | X.X | xxx | XXX. | xx | xx |
| | Day 3 | xxxx-xx-xxTxxx.xx(x) | .XXX L | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Day 7 | xxxx-xx-xxTxxx.xx(x) | XXX. | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Day 20 | xxx-xx-xxTxx | XXX. | XXX | X.XX | X.X | XXX | XXX. | XX | XX |
| | Day 21 | xxx-xx-xxTxx | .xxx L | xxx | X.XX | x.x | xxx | XXX. | XX | xx |
| | Day 22 | xxxx-xx-xxTxx:xx (xx) | .xxx L | XXX | X.XX | X.X | XXX | XXX. | xx | XX |

H=High, L=Low, ET=Early Termination.

HCT = Hematocrit; HGB = Hemoglobin; RBC = Erythrocytes; WBC=Leukocytes; PLAT = Platelets, RETI=Reticulocytes, aPTT2=Activated partial thromboplastin time, PT2=Prothrombin time.

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX

[Programming Note: For out of range results, use bold font and superscript L or H as shown in the example]

Protocol No. TBAJ-876-CL002 TKL No. P1980322 TB Alliance

| TB Alliance | |
|---|---|
| Protocol Number: TBAJ-876-CL002 | |
| Listing 16.2.8.4.2: Clinical Laboratory Test Results, Differential Blood Count | lood Count |
| Safety Population | |

| | | | NEUT | TU | LYM | M | MONO | NO. | EOS | S | BASO | 08 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Subject Time Point | Date-Time (Day) | $(10^{4})$ | (Ratio) | $(10^{4})$ | (Ratio) | $(10^{4})$ | (Ratio) | $(10^{4})$ | (Ratio) | $(10^{4})$ | (Ratio) |
| XXX | Screening | xxxx-xx-xxTxx:xx (-xx) | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Day -1 | (x-) $xx:xxTxx-xx-xxx$ | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Day 2 | xxxx-xx-xxTxx:xx(x) | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Day 3 | xxxx-xx-xxTxx:xx(x) | X.X | X.XX | X.X | X.XX | x.x L | x.xx L | X.X | X.XX | X.X | X.XX |
| | Day 7 | xxxx-xx-xxTxx:xx(x) | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Day 20 | xxxx-xx-xxTxx:xx (xx) | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Day 21 | xxxx-xx-xxTxx:xx (xx) | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Day 22 | xxxx-xx-xxTxx:xx (xx) | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX | X.X | X.XX |
| | Day 25/ET | xxxx-xx-xxTxx:xx (xx) | X.X | X.XX | X.X | X.XX | X.X | x.xx | X.X | X.XX | X.X | X.XX |

H = High; L = Low; ET=Early Termination.

NEUT = Neutrophils; LYM = Lymphocytes; MONO = Monocytes; EOS = Eosinophils; BASO = Basophils

Generated on XX/XX/XX:XXXX by XXXXXX / Uses: XX

[Programming Note: For out of range results, use bold font and superscript L or H as shown in the example]


| TB Alliance | Page X of Y |
|---|---|
| Flowcol (Millott: TDAJ-9/0-CE002 | Listing 16.2.8.4.3: Clinical Laboratory Test Results, Electrolytes and Renal Function |
| | Safety Population |

| Subject | Subject Time Point | Date-Time (Day) | SODIUM (mmol/L) | K<br>(mmol/L) | CL (mmol/L) | BICARB (mmol/L) | CA<br>(mmol/L) | MG<br>(mmol/L) | UREAN (mmol/L) | CREAT (umol/L) |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Screening | (xx-) xx:xxTxx-xx-xx | XXXX | × | XXX | × | ×× | XXX | ×× | ×× |
| | Day -1 | $(x-)$ $\times \times \times$ | XXXX.X | X.X | XXX | XX | x.x | X.XX | x.x | XX |
| | Day 2 | (x) xx:xxTxx-xx-xxx | XXX.X | x.x | xxx | X | X.X | X.XX | X.X | XX |
| | Day 3 | xxxx-xx-xxTxx | XXX.X | x.x | xxx | X | X.X | X.XX | X.X | XX |
| | Day 7 | xxxx-xx-xxTxx | XXX.X | x.x | xxx | X | X.X | X.XX | X.X | XX |
| | Day 20 | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX.X | X.X | XXX | XX | X.X | X.XX | X.X | XX |
| | Day 21 | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX.X | X.X | XXX | XX | X.X | X.XX | X.X | XX |
| | Day 22 | XXXX-XX-XX = XX = XX = XX = XX = XX = X | XXX.X | X.X | XXX | XX | X.X | X.XX | X.X | XX |
| | Day 25/ET | xxxx-xx-xxTxxxxx | XXXX.X | X.X | XXX | XX | x.x | x.xx | x.x | x |

H=High, L=Low, ET=Early Termination.

K=Potassium, CL=Chloride, BICARB=Bicarbonate, CA=Calcium, MG=Magnesium, UREAN=Urea nitrogen, CREAT=Creatinine

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX

[Programming Note: For out of range results, use bold font and superscript L or H]


| F1010001 | rrotocol number. 1543-870-CL002 | | Listing 16.2.8.4. <sup>∠</sup> | 4: Clinical Laboratory Test<br>Safety Population | Listing 16.2.8.4.4: Clinical Laboratory Test Results, Liver Function Safety Population | Liver Function | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Subject Time Point | Date-Time (Day) | ALT (ukat/L) | AST (ukat/L) | ALP (ukat/L) | TBILI (umol/L) | DBILI (umol/L) | (umol/L) | LDH<br>(ukat/L) |
| XXX | Screening | xxxx-xx-xxTxx:xx (-xx) | X.XX | XX.X | X.XX | X.X | X.X | X.X | X.XX |
| | Day -1 | xxxx-xx-xxTxx:xx (-x) | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Day 2 | xxxx-xx-xxTxx:xx(x) | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Day 3 | xxxx-xx-xxTxx:xx(x) | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Day 7 | xxxx-xx-xxTxx:xx(x) | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Day 20 | xxxxx-xx-xxTxx (xx) | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Day 21 | (xx) xx:xxTxx-xx-xxx | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Day 22 | xxxxxxxxxxxxxxxxxxxxxx | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |
| | Day 25/ET | xxxx-xx-xxxxxx (xx) | X.XX | X.XX | X.XX | X.X | X.X | X.X | X.XX |

H=High, L=Low, ET=Early Termination.
ALT=Alanine transaminase, AST=Aspartate transaminase, ALP=Alkaline phosphatase, TBILI=Total bilirubin, DBILI=Direct bilirubin, IBILI=Indirect bilirubin, LDH=Lactate dehydrogenase.

Generated on XX/XX/XX:XXXX by XXXXXX / Uses: XX

[Programming Note: For out of range results, use bold font and superscript L or H]


| FIOLOGO | riolocol number: 1543-8/0-CL002 | ·o/o-c.cu02 | ing 16.2.8.4.5: C | 16.2.8.4.5: Clinical Laboratory Test Results, Other Serum Chemistry Safety Population | 'est Results, Oth<br>ulation | ıer Serum Chemistr | >- | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Subject Time Point | Date-Time (Day) | TPROT (g/L) | GLUC (mmol/L) | ALB<br>(g/L) | URAC<br>(umol/L) | CPK (ukat/L) | AMY<br>(ukat/L) | LIP<br>(ukat/L) |
| XXX | Screening | xxxx-xx-xxTxx:xx (-xx) | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day -1 | (x-) xx:xxTxx-xx-xxx | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day 2 | xxxx-xx-xxTxx:xx(x) | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day 3 | xxxx-xx-xxTxx:xx (x) | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day 7 | xxxx-xx-xxTxx | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day 20 | xxxx-xx-xxTxx:xx (xx) | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day 21 | xxxx-xx-xxTxx:xx (xx) | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day 22 | (xx) xx:xxTxx-xx-xxx | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| | Day 25/ET | XXXX-XX-XXTXX:XX (XX) | XX | XXX | XX | XXX | X.XX | X.XX | X.XX |
| H=High,<br>TPROT= | H=High, L=Low, ET=Early Termination. TPROT=Total protein, GLUC=Glucose, / | H=High, L=Low, ET=Early Termination. TPROT=Total protein, GLUC=Glucose, ALB=Albumin, URAC=Uric acid, CPK=Creatinine phosphokinase, AMY=Amylase, LIP=Lipase | 1, URAC=Uric a | cid, CPK=Creatinin | e phosphokinas | e, AMY=Amylase, | LIP=Lipase | | |
| Storogo | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | VY - 2001 I / VYVVV VXVVV VV VV VV VV VV VV VV | ^^ | | | | | | |
| Collegan | CO OT クク/クク/ク | A.AAAA UV AAAAA / USES. | VV | | | | | | |

[Programming Note: For out of range results, use bold font and superscript L or H]


| TB Alliance Protocol Nur | TB Alliance Protocol Number: TBAJ-876-CL002 | -876-CL002 | | | | | | | Page X of Y |
|---|---|---|---|---|---|---|---|---|---|
| | | | isting 16.2.8. | Listing 16.2.8.4.6: Clinical Laboratory Test Results, Urinalysis, Part 1 Safety Population | ory Test Results, Upulation | Jrinalysis, Part 1 | | | |
| Subject | Time<br>Point | Date-Time (Day) | hd | SpG (g/mL) | GLUC | KET | BILI | CREAT | SOD |
| XXX | Screening | xxxx-xx-xxTxx:xx (-xx) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| | Day -1 | (x-) xx:xxTxx-xx-xxx | X.X | X.XXX | xxx | XXX | XXX | XXX | XXX |
| | Day 2 | xxxx-xx-xxTxxx.xx(x) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 3 | xxxx-xx-xxTxx:xx(x) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 7 | xxxx-xx-xxTxx:xx(x) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 20 | xxxx-xx-xxTxx:xx (xx) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 21 | xxxx-xx-xxTxx:xx (xx) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 22 | xxxx-xx-xxTxx:xx (xx) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 25/ET | xxxx-xx-xxTxx:xx (xx) | X.X | X.XXX | XXX | XXX | XXX | XXX | XXX |
| A=Abnor<br>SpG=Spe | A=Abnormal, ET=Early Termination.<br>SpG=Specific gravity, GLUC=Glucos | A=Abnormal, ET=Early Termination. SpG=Specific gravity, GLUC=Glucose, KET=Ketones, l | BILI=Bilirub | BILI=Bilirubin, CREAT=Creatinine, SOD=Sodium. | ne, SOD=Sodium | | | | |

[Programming Note: For out of range results, use bold font and superscript A.]

Protocol No. TBAJ-876-CL002 TKL No. P1980322 TB Alliance

TB Alliance
Protocol Number: TBAJ-876-CL002

Listing 16.2.8.4.7: Clinical Laboratory Test Results, Urinalysis, Part 2 Safety Population

| Microscopic Examination (if indicated) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| LEUK | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| NIT | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| OCC | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| PROT | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Date-Time (Day) | (xx-) xx:xxTxx-xx-xxx | (x-) $XX:XX TXX-XX-XXX$ | xxxx-xx-xxTxxx (x) | XXXX-XX-XX = XXX | XXXX-XX-XX = XXX | xxxx-xx-xxTxx:xx(xx) | xxxx-xx-xxTxx:xx(xx) | xxxx-xx-xxTxx:xx(xx) | xxxx-xx-xxTxx:xx (xx) |
| Subject Time Point | Screening | Day -1 | Day 2 | Day 3 | Day 7 | Day 20 | Day 21 | Day 22 | Day 25/ET |
| Subject | XXX | | | | | | | | |

A=Abnormal, ET=Early Termination. PROT=Protein, OCC=Occult blood, NIT=Nitrite, LEUK=Leukocyte esterase.

**TB Alliance**Protocol Number: TBAJ-876-CL002

Listing 16.2.8.4.8: Laboratory Values Outside of Normal Range

Safety Population

| nplect | Time Point | Subject Time Point Date-Time (Day) | Panel | Parameter (Unit) | Reference Range Result | Result | Abnormality |
|---|---|---|---|---|---|---|---|
| XXX | Day -1 | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Chemistry | XXXXXX (XX) | XXXX, XXXX | XX.XX | Low |
| | Day 7 | xxxxx-xx-xxTxx:xx (x) | Chemistry | XXXXXX (XX) | XXXX, XXXX | XX.XX | Low |
| XXX | Day 22 | (x-) xx:xxTxx-xx | Hematology | (xx) xxxxxx | XXXX, XXXX | XX.XX | High |

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

[Programming Note: Use SDTM terms for parameter and unit.]

| Day 25 / Early Termination | Check-in (Day -1) | Screening | |
|---|---|---|---|
| | l and Serum Pregnancy Test Results<br>ulation | Listing 16.2.8.5: Childbearing Potential and Serum Pregnancy Test Results Safety Population | |
| Page X of Y | | | TB Alliance<br>Protocol Number: TBAJ-876-CL002 |

| | | Screening | | Check-in (Day -1) | y -1) | Day 25 / Early Termination | rmination |
|---|---|---|---|---|---|---|---|
| Subject | Subject Childbearing Potential | Date-Time | Result | Date-Time | Result | Date-Time | Result |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxx-xx-xxTxx:xx (-x) | XXXXXXXXX | xxxx-xx-xxTxx.xx (-x) | XXXXXXXXX | xxxx-xx-xxTxx:xx (-x) xxxxxxxxxxx | XXXXXXXXXX |
| XXX | XXXXXXXXXXXXXXXXXXXX | (x-) xx:xxTxx-xx-xxxx | XXXXXXXXX | xxxxxxxxxx (x-) xx:xxTxx-xxx | XXXXXXXXXX | xxxxxxxxxx (-x) xxxxxxxxxxx | XXXXXXXXX |
| XXX | xxxxxxxxxxxxxxxxxx (FSH= xxx) | xxxx-xx-xxTxx:xx (-x) | XXXXXXXXX | (x-) xx:xxTxx-xx-xx | XXXXXXXXXX | XXXXXXXXXX (-x) XX:XXTXX-XX-XX-XXXXXXXXX (-x) XX:XXTXX-XX-XXXXX | XXXXXXXXX |
| XXX | XXXXXXXXXXXXXX | xxxxxxxxxx (-x) xxxxxxxxxx | XXXXXXXXX | (x-) xx:xxTxx-xx-xxxx | XXXXXXXXXX | XXXX-XX-XX-XXTXX:XX (-x) XXXXXXXXXXX XXXX-XX-XX-XXXTXX:XX (-x) | XXXXXXXXX |

Note: Include serum FSH test result as shown for those subjects who present data.


| TB Alliance Protocol Number | TB Alliance<br>Protocol Number: TBAJ-876-CL002 | Page X of Y |
|---|---|---|
| | | Listing 16.2.9: General Comments Safety Population |
| Subject | Comment Reference | Comment |
| XXX | XXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Generated on X | Generated on XX/XX/XX:XXXX by XXXX / Uses: CO | //uses: CO |